CLINICAL TRIAL: NCT02422797
Title: A Phase III, Randomized, Multicenter, Parallel-group, Non-inferiority Study Evaluating the Efficacy, Safety, and Tolerability of Switching to Dolutegravir Plus Rilpivirine From Current INI-, NNRTI-, or PI-based Antiretroviral Regimen in HIV-1-infected Adults Who Are Virologically Suppressed
Brief Title: Regimen Switch to Dolutegravir + Rilpivirine From Current Antiretroviral Regimen in Human Immunodeficiency Virus Type 1 Infected and Virologically Suppressed Adults (SWORD-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201637; 2014-005148-16 (EudraCT Number)
Record Dates: First submitted 2015-04-09; First posted 2015-04-21 (Estimated); Results first posted 2017-10-24 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
Keywords: HIV; NNRTI-sparing; two-drug regimen; nucleoside reverse transcriptase inhibitors; protease inhibitor; integrase inhibitor; non-nucleoside reverse transcriptase inhibitor; dolutegravir plus rilpivirine; virologically-suppressed
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Current antiretroviral regimen (CAR) (Active Comparator): Participants continued to receive their current antiretroviral regimen (two nucleoside reverse transcriptase inhibitor [NRTIs] + a third agent). A third agent included either an: integrase strand transfer inhibitor (INSTI), a non-nucleoside reverse transcriptase inhibitor (NNRTI) or a protease inhibitor (PI). CAR was administered according to the approved labeling in an open-label fashion up to Week 52 during early switch phase. At Week 52, participants with human immunodeficiency virus-1 (HIV-1) ribonucleic acid (RNA) <50 copies per milliliter (c/mL), switched to DTG 50 mg + RPV 25 mg once daily and were followed-up through the Late Switch Phase, at Week 148 and through the Continuation Phase, after Week 148.
  Interventions: Drug: CAR
- DTG + RPV (Experimental): Participants received DTG 50 milligrams (mg) + RPV 25 mg together once daily at approximately the same time, with a meal, in an open-label fashion up to Week 52 during early switch phase. Participants continued to receive DTG 50 mg + RPV 25 mg up to Week 148 during the Late Switch Phase.
  Participants who successfully completed 148 weeks of treatment were given the opportunity to continue to receive DTG + RPV once daily in the Continuation Phase (after Week 148).
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg

INTERVENTIONS:
Drug: DTG 50 mg — Participants received one oral tablet of 50 mg DTG daily administered concomitantly with RPV. Each DTG tablet contained 52.62 mg dolutegravir sodium salt, which was equivalent to 50 mg dolutegravir free acid.
  Arms: DTG + RPV
Drug: RPV 25 mg — Participants received DTG 50 milligrams (mg) + RPV 25 mg together once daily at approximately the same time, with a meal, in an open-label fashion up to Week 52 during early switch phase. Participants continued to receive DTG 50 mg + RPV 25 mg up to Week 148 during the Late Switch Phase.
  Participants who successfully completed 148 weeks of treatment were given the opportunity to continue to receive DTG + RPV once daily in the Continuation Phase (after Week 148), one oral tablet of 25 mg RPV daily administered concomitantly with DTG along with a meal. Each RPV tablet contained 27.5 mg of rilpivirine hydrochloride, which was equivalent to 25 mg of RPV.
  Arms: DTG + RPV
Drug: CAR — CAR included the following combinations: 2 NRTIs + 1 INI, 2 NRTIs + 1 NNRTI, or 2 NRTIs + 1 PI.
  Arms: Current antiretroviral regimen (CAR)

SUMMARY:
The aim of this study was to determine if virologically suppressed, human immunodeficiency virus type 1 (HIV-1) infected adults on an antiretroviral regimen (including 2 nucleoside reverse transcriptase inhibitors [NRTIs] plus a third agent) remain suppressed upon switching to a two-drug regimen with dolutegravir (DTG) + rilpivirine (RPV). The study primarily assessed the non-inferiority antiviral activity of switching to DTG + RPV once daily compared to the continuation of current antiretroviral regimen (CAR) up to Week 48 with a switch visit for eligible subjects in the CAR group to initiate DTG + RPV therapy at Week 52. CAR included 2 NRTIs plus 1 HIV-1 integrase inhibitor (INI), or 1 non-nucleoside reverse transcriptase inhibitor (NNRTI), or 1 protease inhibitor (PI). The study included a 148-week open-label treatment phase, comprising of an Early Switch Phase (Day 1 to Week 52) and a Late Switch Phase (Week 52 to Week 148). The participants fulfilling the study eligibility criteria participated in the Early Switch Phase where they either switched from their CAR to DTG + RPV, or continued taking their CAR, until Week 52. At the end of Early Switch Phase, eligible participants proceeded to the Late Switch Phase where all participants in both DTG + RPV and CAR treatment groups received DTG + RPV therapy until Week 148. After Week 148, subjects could have been eligible to continue to receive DTG +RPV in the Continuation Phase.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been able to understand and comply with protocol requirements, instructions, and restrictions.
* Participants must have been likely to complete the study as planned.
* Participants must have been considered appropriate candidates for participation in an investigative clinical trial with oral medication (e.g., no active substance abuse, acute major organ disease, or planned long-term work assignments out of the country, etc.).
* HIV-1 infected men or women of greater than or equal to (>=)18 years of age.
* Must have been on uninterrupted current regimen (either the initial or second combination antiretroviral therapy [cART] regimen) for at least 6 months prior to screening; Any prior switch, defined as a change of a single drug or multiple drugs simultaneously, must have occurred due to tolerability and/or safety concerns or access to medications, or convenience/simplification. Acceptable stable cART regimens prior to screening include 2 NRTIs plus INI (either the initial or second cART regimen), or an NNRTI (either the initial or second cART regimen), or a Boosted PI (or atazanavir unboosted) (either the initial or second PI-based cART regimen).
* Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: one within the 6 to 12 month window, and one within 6 months prior to Screening;
* Plasma HIV-1 RNA <50 c/mL at Screening;
* A female may have been eligible to enter and participate in the study if she was of : Non-child-bearing potential either defined as post-menopausal (12 months of spontaneous amenorrhea and >=45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or, Child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy: Complete abstinence from intercourse from 2 weeks prior to administration of study drug, throughout the study, and for at least 2 weeks after discontinuation of all study medications and completion of the Follow-up visit; Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion); Male partner sterilization with documentation of azoospermia prior to the female participant's entry into the study and this male is the sole partner for that participant; The documentation on male sterility could come from the site personnel's review of participant's medical records, medical examination, and/or semen analysis, or medical history interview provided by her or her partner; Approved hormonal contraception for participants randomly assigned to DTG + RPV arm (and for participants randomly assigned to CAR following switch to DTG + RPV at Week 52) or approved hormonal contraception plus a barrier method for participants assigned to CAR through Week 52; Approved hormonal contraception included: Combined estrogen and progestogen oral contraceptive, Contraceptive subdermal implant, Injectable progestogen, Contraceptive vaginal ring, Percutaneous contraceptive patches. Any other method with published data showing that the expected failure rate is <1% per year. Any contraception method must have been used consistently, in accordance with the approved product label during treatment with study drug and for at least 2 weeks after discontinuation of study drug and completion of the Follow-Up Visit. The investigator was responsible for ensuring that participants understand how to properly use these methods of contraception. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal were not acceptable methods of contraception.
* Participants who were willing and able to understand requirements of study participation and provided signed and dated written informed consent prior to screening.
* For participants enrolled in France: participants were eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

Exclusionary Criteria prior to screening or Day 1:

* Within 6 months prior to Screening and after confirmed suppression to <50 c/mL on current ART regimen, any plasma HIV-1 RNA measurement >=50 c/mL.
* Within the 6 to 12 month window prior to screening and after confirmed suppression to <50 c/mL, any plasma HIV-1 RNA measurement >200 c/mL.
* Within the 6 to 12 month window prior to screening and after confirmed suppression to <50 c/mL, 2 or more plasma HIV-1 RNA measurements >=50 c/mL.
* Any drug holiday during the window between initiating first HIV ART and 6 months prior to screening, except for brief periods (less than 1 month) where all ART was stopped due to tolerability and/or safety concerns.
* Any switch to a second line regimen, defined as change of a single drug or multiple drugs simultaneously, due to virologic failure to therapy (defined as a confirmed plasma HIV 1 RNA measurement >=400 c/mL after initial suppression to <50 c/mL while on first line HIV therapy regimen).

Exclusionary medical conditions:

* Women who were pregnant, breastfeeding or planned to become pregnant or breastfeed during the study.
* Any evidence of an active Centers for Disease Control and Prevention Category C disease. Exceptions included cutaneous Kaposi's sarcoma not requiring systemic therapy and historic CD4+ lymphocyte counts of <200 cells per cubic millimeter (cells/mm^3).
* Participants with severe hepatic impairment (Class C) as determined by Child-Pugh Classification.
* Unstable liver disease (as defined by the presence of any of the following: ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), and Hepatitis B surface antibody (HBsAb) as follows: Participants positive for HBsAg were excluded; Participants positive for anti-HBc (negative HBsAg status) and negative for HBsAb were excluded.
* Participants with an anticipated need for any Hepatitis C virus (HCV) therapy during the Early Switch Phase and for interferon-based therapy for HCV throughout the entire study period.
* History or presence of allergy to the study drugs or their components or drugs of their class;
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the participant prior to randomization;
* Participants who in the investigator's judgment posed a significant suicidality risk. Participant's history of suicidal behavior and/or suicidal ideation should have been considered when evaluating for suicide risk;
* Any pre-existing physical or mental condition which, in the opinion of the Investigator, could have interfered with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which could have compromised the safety of the participants;
* Any condition which, in the opinion of the Investigator, could have interfered with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to take oral medication;

Exclusionary Treatments prior to Screening or Day 1:

* Use of medications which were associated with Torsades de Pointes.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Treatment with any of the following agents within 28 days of Screening: radiation therapy; cytotoxic chemotherapeutic agents; any immunomodulators that alter immune responses.
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to Day 1 of this study.
* Participants who were participating or anticipated to be selected to participate in any other interventional study, with the exception of the DEXA sub-study 202094, after randomization
* A history of use of any regimen consisting of only single NNRTI therapy (even if only for peri-partum treatment), or only single or dual NRTI therapy prior to starting cART.
* Current or prior history of etravirine (ETR) use.
* Current use of tipranavir/ritonavir or fosamprenavir/ritonavir.
* Participants receiving any prohibited medication and who were unwilling or unable to switch to an alternate medication.

Exclusionary Laboratory Values or Clinical Assessments at Screening:

* Evidence of viral resistance based on the presence of any resistance associated major PI, INI, NRTI, or NNRTI mutation and integrase (IN) resistance associated substitution R263K in any available prior resistance genotype assay results.
* Any verified Grade 4 laboratory abnormality, with the exception of Grade 4 lipid abnormalities. A single repeat test was allowed during the Screening period to verify a result.
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's participation in the study of an investigational compound.
* Alanine aminotransferase (ALT) >=5 × upper limit of normal (ULN), or ALT >=3 × ULN and bilirubin >=1.5 × ULN (with greater than [>] 35% direct bilirubin).
* Corrected QT interval (QTc [Bazett]) >450 milliseconds or QTc (Bazett) >480 milliseconds for participants with bundle branch block. The QTc was the QT interval corrected for heart rate according to Bazett's formula (QTcB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (52):
- United States (12):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Buffalo, Texas
  - GSK Investigational Site, Seattle, Washington
- Argentina (2):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Rosario
- Australia (2):
  - GSK Investigational Site, Darlinghurst
  - GSK Investigational Site, Sydney
- Canada (4):
  - GSK Investigational Site, Montreal
  - GSK Investigational Site, Regina
  - GSK Investigational Site, Toronto
  - GSK Investigational Site, Vancouver
- France (6):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Denis
  - GSK Investigational Site, Tourcoing
- Germany (4):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Hanover
- Italy (2):
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Milan
- Russia (4):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
- Spain (12):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cartagena
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Santa Cruz La Laguna
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
- Taiwan (3):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, New Taipei City
  - GSK Investigational Site, Taichung
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Llibre JM, Hung CC, Brinson C, et al. Efficacy, safety, and tolerability of dolutegravir plus rilpivirine for the maintenance of virologic suppression in HIV-1-infected adults: the phase III, randomized, open-label, active-controlled, noninferiority SWORD-1 and SWORD-2 studies. Lancet [epublished ahead of print] 6 January 2018.
- [Derived] Aboud M, Orkin C, Podzamczer D, Bogner JR, Baker D, Khuong-Josses MA, Parks D, Angelis K, Kahl LP, Blair EA, Adkison K, Underwood M, Matthews JE, Wynne B, Vandermeulen K, Gartland M, Smith K. Efficacy and safety of dolutegravir-rilpivirine for maintenance of virological suppression in adults with HIV-1: 100-week data from the randomised, open-label, phase 3 SWORD-1 and SWORD-2 studies. Lancet HIV. 2019 Sep;6(9):e576-e587. doi: 10.1016/S2352-3018(19)30149-3. Epub 2019 Jul 12. PMID 31307948
- [Derived] Llibre JM, Hung CC, Brinson C, Castelli F, Girard PM, Kahl LP, Blair EA, Angelis K, Wynne B, Vandermeulen K, Underwood M, Smith K, Gartland M, Aboud M. Efficacy, safety, and tolerability of dolutegravir-rilpivirine for the maintenance of virological suppression in adults with HIV-1: phase 3, randomised, non-inferiority SWORD-1 and SWORD-2 studies. Lancet. 2018 Mar 3;391(10123):839-849. doi: 10.1016/S0140-6736(17)33095-7. Epub 2018 Jan 6. PMID 29310899
- [Derived] McComsey GA, Lupo S, Parks D, Poggio MC, De Wet J, Kahl LP, Angelis K, Wynne B, Vandermeulen K, Gartland M, Cupo M, Aboud M; 202094 Sub-Study Investigators. Switch from tenofovir disoproxil fumarate combination to dolutegravir with rilpivirine improves parameters of bone health. AIDS. 2018 Feb 20;32(4):477-485. doi: 10.1097/QAD.0000000000001725. PMID 29239893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 60 centers in 11 countries.
Pre-assignment Details: 518 participants were randomized and 2 participants withdrew before being exposed to study drug. The study included an Early Switch Phase, a Late Switch Phase, and a Continuation Phase.
Period: Early Switch Phase (Up to Week 52)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Started | 261 | 255
Completed | 245 | 239
Not Completed | 16 | 16
Not completed — Adverse Event | 11 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 3
Not completed — Reached stopping criteria | 1 | 1
Not completed — Withdrawal by Subject | 2 | 7
Period: Late Switch Phase (Week 52 to Week 148)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Started | 245 | 239
Completed | 222 | 221
Not Completed | 23 | 18
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 10 | 6
Not completed — Lack of Efficacy | 5 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Reached stopping criteria | 1 | 0
Not completed — Protocol Violation | 3 | 0
Period: Continuation Phase(Week 148 to Week 410)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Started | 208 | 204
Completed | 201 | 194
Not Completed | 7 | 10
Not completed — Investigator discretion | 1 | 2
Not completed — Lost to Follow-up | 0 | 3
Not completed — Subject reached protocol-defined stopping criteria | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR) | Total
Number analyzed (Participants) | 261 | 255 | 516
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.3 (11.34) | 43.2 (9.64) | 43.3 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 57 | 119
  Male | 199 | 198 | 397
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 7 | 18
  Central/South Asian Heritage | 0 | 1 | 1
  Japanese/East Asian (EA) Heritage (H.)/South EA H. | 13 | 15 | 28
  Black/African American | 13 | 19 | 32
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White | 223 | 212 | 435
  African American/ African H. and White | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 48 Using Snapshot Algorithm
Description: Percentage of participants with plasma HIV 1 RNA < 50 c/mL at Week 48 using the Food and Drug Administration (FDA) snapshot algorithm was assessed to demonstrate the non-inferior antiviral activity of switching to DTG+RPV once daily compared to continuation of CAR over 48 weeks in HIV-1 infected antiretroviral therapy (ART)-experienced participants. Virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment within the window of the visit of interest. Plasma samples were collected for quantitative analysis of HIV-1 RNA.
Time Frame: Week 48
Population: The Analysis was performed on the Intent-to-Treat Exposed (ITT-E) population which consisted of all randomly assigned participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Percentage of participants | 94 | 94
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Non-Inferiority — Non-inferiority was concluded if the lower bound of a two-sided 95% confidence interval for the difference in response rates between the two treatment arms was greater than -10%; Risk Difference (RD) = 0.2, 95% CI 2-sided [-3.9 to 4.2] — Estimates based on Cochran-Mantel Haenszel stratified analysis adjusting for Baseline stratification factors: Age group (< or >=50 years old) and Baseline third agent (PI, NNRTI, INSTI)

2. Secondary Outcome: Changes From Baseline in Cluster Designation (CD)4+ Lymphocyte Count at Weeks 24 and 48
Description: Blood samples were collected and CD4+ cell count assessment by flow cytometry was carried out to evaluate the immunological activity of DTG + RPV once daily compared to continuation of CAR. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Weeks 24 and 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per millimeter cube (mm^3)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Cells per millimeter cube (mm^3)
  Week 24: number analyzed (Participants) | 251 | 250
  Week 24 | 42.0 (172.29) | 42.4 (164.85)
  Week 48: number analyzed (Participants) | 245 | 241
  Week 48 | 28.0 (169.35) | 18.4 (159.34)

3. Secondary Outcome: Percentage of Participants With Plasma HIV 1 RNA <50 c/mL at Week 24 Using Snapshot Algorithm
Description: Percentage of participants with plasma HIV 1 RNA <50 c/mL at Week 24 using the FDA snapshot algorithm was assessed to evaluate the antiviral activity of DTG +RPV once daily compared to continuation of CAR. Virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment within the window of the visit of interest. Plasma samples were collected for quantitative analysis of HIV-1 RNA.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Percentage of participants | 97 | 98
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; Risk Difference (RD) = -1.1, 95% CI 2-sided [-4.0 to 1.8] — Cochran-Mantel Haenszel stratified analysis adjusting for Baseline stratification factors: Age group (< or >=50 years old) and Baseline third agent (PI, NNRTI, INSTI). No formal non-inferiority margin has been pre-specified for secondary endpoints

4. Secondary Outcome: Number of Participants With Common Non-serious Adverse Event (AE), Any Serious AE (SAE), AE of Maximum Toxicity Grade 1, 2, 3 or 4 and AE Leading to Discontinuation (AELD)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with use of a medicinal product, whether or not considered related to medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention were categorized as SAE. AEs were graded using the Division of Acquired Immunodeficiency Syndrome (DAIDS) grading. Grade 1=mild; Grade 2=moderate, Grade 3=severe and Grade 4=potentially life-threatening. Common AEs were those with >5% incidence for either treatment.
Time Frame: Up to Week 410 or study discontinuation
Population: Safety Population included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 239
Participants
  Common non-serious AE | 166 | 132
  Any SAE | 50 | 32
  Maximum toxicity Grade 1 AE | 78 | 85
  Maximum toxicity Grade 2 AE | 104 | 95
  Maximum toxicity Grade 3 AE | 33 | 29
  Maximum toxicity Grade 4 AE | 13 | 11
  AELD | 23 | 8

5. Secondary Outcome: Number of Participants With Maximum Post-baseline Emergent Chemistry Toxicities Over 48 Weeks
Description: Blood samples were collected to evaluate alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), total bilirubin, chloride, creatinine, glucose, potassium, phosphate, sodium, blood urea nitrogen (BUN), total carbon dioxide, lipase, creatine phosphokinase and creatinine clearance. Value obtained at Day 1 was considered as Baseline value. Number of participants who experienced maximum grade toxicity post-baseline in clinical chemistry over 48 weeks was summarized. Clinical chemistry toxicities were graded using the Division of AIDS Table for Grading Severity of Adult and Pediatric Adverse Events. Grade 1=mild; Grade 2=moderate, Grade 3=severe and Grade 4=potentially life-threatening. For all laboratory parameters, one assessment out of range was sufficient to be considered a chemistry toxicity.
Time Frame: Up to 48 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Participants
  Grade 1 | 92 | 80
  Grade 2 | 72 | 79
  Grade 3 | 11 | 16
  Grade 4 | 1 | 10

6. Secondary Outcome: Number of Participants With Maximum Post-baseline Emergent Hematology Toxicities Over 48 Weeks
Description: Blood samples were collected to evaluate hemoglobin, hematocrit, basophils, eosinophils, lymphocytes, monocytes, neutrophils, mean corpuscular volume (MCV), red blood cell (RBC) count, white blood cell (WBC) count and platelet count. Value obtained at Day 1 was considered as Baseline value. Number of participants who experienced maximum grade toxicity post-baseline in hematology over 48 weeks was summarized. Hematology toxicities were graded using the Division of AIDS Table for Grading Severity of Adult and Pediatric Adverse Events. Grade 1=mild; Grade 2=moderate, Grade 3=severe and Grade 4=potentially life-threatening. For all laboratory parameters, one assessment out of range was sufficient to be considered a hematology toxicity.
Time Frame: Up to 48 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Participants
  Grade 1 | 11 | 11
  Grade 2 | 2 | 2
  Grade 3 | 3 | 0
  Grade 4 | 1 | 0

7. Secondary Outcome: Mean Change From Baseline in High-sensitivity C-reactive Protein (Hs-CRP) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess hs-CRP. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/Liter (L)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 246 | 239
mg/Liter (L) | 0.10 (5.383) | 0.80 (8.527)

8. Secondary Outcome: Mean Change From Baseline in Cystatin C at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess cystatin C. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 246 | 237
mg/L | -0.02 (0.110) | -0.01 (0.108)

9. Secondary Outcome: Mean Change From Baseline in D-Dimer at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess D-Dimer. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomole/L fibrinogen equivalent units
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 239 | 228
Nanomole/L fibrinogen equivalent units | 0.01 (1.629) | -0.13 (2.932)

10. Secondary Outcome: Mean Change From Baseline in Fatty Acid Binding Protein 2 (FABP) and Soluble CD14 at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess FABP and soluble CD14. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Nanogram/milliliter
  FABP: number analyzed (Participants) | 245 | 236
  FABP | -1.50 (1.278) | -0.99 (1.441)
  Soluble CD14: number analyzed (Participants) | 245 | 237
  Soluble CD14 | 456.69 (731.833) | 802.26 (878.304)

11. Secondary Outcome: Mean Change From Baseline in Soluble CD163 and Oxidized Low Density Lipoprotein (LDL) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess soluble CD163 and oxidized LDL. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram(µg)/Liter
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Microgram(µg)/Liter
  Soluble CD163: number analyzed (Participants) | 245 | 236
  Soluble CD163 | 65.38 (180.869) | 53.94 (215.621)
  Oxidized LDL: number analyzed (Participants) | 245 | 237
  Oxidized LDL | 60.87 (504.345) | 13.92 (575.305)

12. Secondary Outcome: Mean Change From Baseline in Retinol Binding Protein (RBP), Serum Creatinine and Glucose at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess RBP, serum creatinine and glucose. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/deciliter (dL)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
mg/deciliter (dL)
  RBP: number analyzed (Participants) | 245 | 237
  RBP | -0.13 (0.825) | 0.00 (0.872)
  Serum creatinine: number analyzed (Participants) | 245 | 241
  Serum creatinine | 0.100 (0.1053) | -0.003 (0.0847)
  Glucose: number analyzed (Participants) | 242 | 235
  Glucose | 0.187 (19.5808) | 3.220 (10.0987)

13. Secondary Outcome: Mean Change From Baseline in Urine Phosphate at Week 48
Description: Urine biomarker samples were collected to at Baseline (Day 1) and Week 48 to assess urine phosphate. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles (mmol)/L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 235 | 229
Millimoles (mmol)/L | 1.335 (16.7211) | -0.798 (15.3771)

14. Secondary Outcome: Mean Change From Baseline in Beta-2-microglobulin (B2M) (Blood and Urine), Urine RBP and 25 Hydroxy-vitamin D (Blood) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess B2M and 25 hydroxy-vitamin D. Urine biomarker samples were collected to assess B2M and RBP. Change from Baseline was calculated as value at indicated time point minus Baseline value. For 25 hydroxy-vitamin D, analysis of changes from Baseline was performed on log-transformed data. Results were transformed back via exponential transformation such that treatment comparisons are assessed via odds ratios.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomoles (nmol)/L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Nanomoles (nmol)/L
  B2M, blood: number analyzed (Participants) | 245 | 238
  B2M, blood | -16.8800 (34.89330) | -4.7501 (43.04355)
  25 hydroxy-vitamin D, blood: number analyzed (Participants) | 243 | 239
  25 hydroxy-vitamin D, blood | -13.9 (25.30) | -9.2 (19.55)
  Urine B2M: number analyzed (Participants) | 72 | 78
  Urine B2M | -173.2820 (1311.24142) | 62.3209 (391.32049)
  Urine RBP: number analyzed (Participants) | 232 | 224
  Urine RBP | -6.8123 (24.09650) | -0.0631 (11.99886)
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.007, ANCOVA — P-value for interaction between treatment group and Baseline third agent (25 hydroxy-vitamin D)
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.011, ANCOVA — P value assessed the difference between treatment groups (25 hydroxy-vitamin D - INSTI); Odds Ratio (OR) = 0.861, 95% CI 2-sided [0.767 to 0.967] — Estimates were calculated from an ANCOVA model adjusting for Baseline third agent class, age, sex, BMI category, smoking status and Baseline biomarker level
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.745, ANCOVA — P value assessed the difference between treatment groups (25 hydroxy-vitamin D - NNRTI); Odds Ratio (OR) = 1.012, 95% CI 2-sided [0.943 to 1.085] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.018, ANCOVA — P value assessed the difference between treatment groups (25 hydroxy-vitamin D - PI); Odds Ratio (OR) = 0.877, 95% CI 2-sided [0.787 to 0.977] — [estimate comment as in outcome 14, analysis 2]

15. Secondary Outcome: Mean Change From Baseline in Urine Albumin/Creatinine Ratio and Urine Protein/Creatinine Ratio at Week 48
Description: Urine biomarker samples were collected at Baseline (Day 1) and Week 48 to assess urine albumin/creatinine ratio and urine protein/creatinine ratio. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams (g)/mol
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Grams (g)/mol
  Urine albumin/creatinine ratio: number analyzed (Participants) | 178 | 181
  Urine albumin/creatinine ratio | -0.78 (5.116) | -0.64 (9.538)
  Urine protein/creatinine ratio: number analyzed (Participants) | 192 | 193
  Urine protein/creatinine ratio | -2.73 (12.683) | 1.23 (5.088)

16. Secondary Outcome: Mean Change From Baseline in Bone-specific Alkaline Phosphatase, Procollagen 1 N-terminal Propeptide, Osteocalcin, Type 1 Collagen C-telopeptides and Soluble Vascular Cell Adhesion Molecule (sVCAM) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess bone-specific alkaline phosphatase, procollagen 1 N-terminal propeptide, osteocalcin, Type 1 Collagen C-telopeptides and sVCAM. Change from Baseline was calculated as value at indicated time point minus Baseline value. For bone-specific alkaline phosphatase, procollagen 1-N-propeptide, osteocalcin and type 1 collagen C-telopeptide, analyses of changes from Baseline were performed on log-transformed data. Results were transformed back via exponential transformation such that treatment comparisons are assessed via odds ratios.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram (ug)/L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Microgram (ug)/L
  Bone-specific alkaline phosphatase: number analyzed (Participants) | 246 | 236
  Bone-specific alkaline phosphatase | -3.18 (5.678) | 0.92 (4.634)
  Procollagen type 1 N-propeptide: number analyzed (Participants) | 245 | 237
  Procollagen type 1 N-propeptide | -5.8 (20.00) | 0.3 (19.28)
  Osteocalcin: number analyzed (Participants) | 245 | 235
  Osteocalcin | -5.11 (7.334) | -1.14 (6.017)
  Type I Collagen C-Telopeptides: number analyzed (Participants) | 243 | 238
  Type I Collagen C-Telopeptides | -0.15 (0.313) | -0.09 (0.344)
  sVCAM: number analyzed (Participants) | 245 | 237
  sVCAM | -2.63 (571.182) | 37.42 (617.486)
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.001, ANCOVA — P-value for interaction between treatment group and Baseline third agent (bone-specific alkaline phosphatase)
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value assessed the difference between treatment groups (bone-specific alkaline phosphatase - NNRTI); Odds Ratio (OR) = 0.728, 95% CI 2-sided [0.686 to 0.773] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.004, ANCOVA — P value assessed the difference between treatment groups (bone-specific alkaline phosphatase - INSTI); Odds Ratio (OR) = 0.865, 95% CI 2-sided [0.785 to 0.954] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value assessed the difference between treatment groups (bone-specific alkaline phosphatase - PI); Odds Ratio (OR) = 0.788, 95% CI 2-sided [0.719 to 0.864] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 5: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.677, ANCOVA — P-value for interaction between treatment group and Baseline third agent (procollagen type 1-N-propeptide)
Statistical Analysis 6: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value assessed the difference between treatment groups (procollagen type 1-N-propeptide); Odds Ratio (OR) = 0.867, 95% CI 2-sided [0.823 to 0.914] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 7: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p < .001, ANCOVA — P-value for interaction between treatment group and Baseline third agent (osteocalcin)
Statistical Analysis 8: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value assessed the difference between treatment groups (osteocalcin - NNRTI); Odds Ratio (OR) = 0.853, 95% CI 2-sided [0.799 to 0.910] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 9: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.028, ANCOVA — P value assessed the difference between treatment groups (osteocalcin - INSTI); Odds Ratio (OR) = 0.886, 95% CI 2-sided [0.796 to 0.987] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 10: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value assessed the difference between treatment groups (osteocalcin - PI); Odds Ratio (OR) = 0.743, 95% CI 2-sided [0.672 to 0.822] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 11: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.782, ANCOVA — P-value for interaction between treatment group and Baseline third agent (type 1 collagen cross-linked C-telopeptide)
Statistical Analysis 12: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value assessed the difference between treatment groups (type 1 collagen cross-linked C-telopeptide); Odds Ratio (OR) = 0.818, 95% CI 2-sided [0.751 to 0.891] — [estimate comment as in outcome 14, analysis 2]

17. Secondary Outcome: Mean Change From Baseline in Interleukin 6 (IL-6) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess IL-6. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms (ng)/L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 245 | 237
Nanograms (ng)/L | -0.08 (2.373) | -0.07 (2.761)

18. Secondary Outcome: Mean Change From Baseline in Insulin Resistance Based on Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess insulin resistance. Change from Baseline was calculated as value at indicated time point minus Baseline value. The homeostatic model assessment (HOMA) of insulin resistance (HOMA-IR ) index , the product of basal glucose and insulin levels divided by 22.5, is regarded as a simple, inexpensive, and reliable surrogate measure of insulin resistance.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: HOMA-IR Score
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 237 | 224
HOMA-IR Score | 0.50 (4.780) | 0.80 (3.938)

19. Secondary Outcome: Mean Change From Baseline in Fasting Lipids at Weeks 24 and 48
Description: Blood samples were collected at Baseline (Day 1), Week 24 and Week 48 to assess fasting lipids which included total cholesterol, low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol and triglycerides. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Weeks 24 and 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles (mmol)/L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Millimoles (mmol)/L
  Total cholesterol, Week 24: number analyzed (Participants) | 237 | 229
  Total cholesterol, Week 24 | -0.015 (0.7539) | 0.020 (0.5777)
  Total cholesterol, Week 48: number analyzed (Participants) | 237 | 230
  Total cholesterol, Week 48 | -0.079 (0.7926) | -0.038 (0.6148)
  LDL cholesterol calculation, Week 24: number analyzed (Participants) | 231 | 221
  LDL cholesterol calculation, Week 24 | 0.085 (0.5940) | 0.055 (0.5232)
  LDL cholesterol calculation, Week 48: number analyzed (Participants) | 229 | 220
  LDL cholesterol calculation, Week 48 | -0.049 (0.6276) | -0.076 (0.5280)
  HDL cholesterol direct, Week 24: number analyzed (Participants) | 237 | 229
  HDL cholesterol direct, Week 24 | -0.024 (0.2365) | -0.051 (0.2258)
  HDL cholesterol direct, Week 48: number analyzed (Participants) | 237 | 230
  HDL cholesterol direct, Week 48 | 0.051 (0.2386) | 0.049 (0.2489)
  Triglycerides, Week 24: number analyzed (Participants) | 237 | 229
  Triglycerides, Week 24 | -0.184 (1.0102) | 0.040 (0.9164)
  Triglycerides, Week 48: number analyzed (Participants) | 237 | 230
  Triglycerides, Week 48 | -0.169 (1.0062) | -0.021 (1.0156)

20. Secondary Outcome: Number of Participants With Genotypic Resistance-Early Switch Phase
Description: Plasma samples were collected for drug resistance testing. Genotypic Resistance data for the following drugs (Rilpivirine [RPV], Dolutegravir [DTG]) in participants Meeting Confirmed Virologic Withdrawal (CVW) criteria has been presented.
Time Frame: Up to Week 48
Population: The analysis was performed on the CVW resistance Population which was comprised of all participants in the ITT-E Population who met CVW through the end of visit window (Week 48, Week 100 or Week 148) and have available on-treatment genotypic resistance data at the time CVW criterion is met.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1 | 0
Participants
  INSTI, DTG, Susceptible | 1 |
  INSTI, DTG, Potential low-level resistance | 0 |
  INSTI, DTG, Low-level resistance | 0 |
  INSTI, DTG, Intermediate resistance | 0 |
  INSTI, DTG, High-level resistance | 0 |
  NNRTI, RPV, Susceptible | 0 |
  NNRTI, RPV, Potential low-level resistance | 0 |
  NNRTI, RPV, Low-level resistance | 0 |
  NNRTI, RPV, Intermediate resistance | 1 |
  NNRTI, RPV, High-level resistance | 0 |

21. Secondary Outcome: Number of Participants With Genotypic Resistance-DTG+RPV Arm Through Early and Late Switch Phase
Description: Plasma samples were collected for drug resistance testing. Genotypic Resistance data for the following drugs (DTG, Elvitegravir [EVG], Raltegravir [RAL], Delavirdine [DLV], Efavirenz [EFV], Etravirine [ETR], Nevirapine [NVP], RPV, Lamivudine [3TC], Abacavir [ABC], FTC, TDF, Zidovudine [ZDV], Stavudine [d4T], Didanosine [ddI], Atazanavir/r [ATV/r], DRV/r, Fosamprenavir/r [FPV/r], Indinavir/r [IDV/r], Lopinavir/r [LPV/r], Nelfinavir [NFV], Ritonavir [RTV], Saquinavir/r [SQV/r], Tipranavir/r [TPV/r]) in participants Meeting Confirmed Virologic Withdrawal Criteria has been presented.
Time Frame: Up to Week 148
Population: CVW resistance Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 2
Participants
  INI, DTG, Susceptible | 2
  INI, DTG, Potential low-level resistance | 0
  INI, DTG, Low-level resistance | 0
  INI, DTG, Intermediate resistance | 0
  INI, DTG, High-level resistance | 0
  INI, EVG, Susceptible | 2
  INI, EVG, Potential low-level resistance | 0
  INI, EVG, Low-level resistance | 0
  INI, EVG, Intermediate resistance | 0
  INI, EVG, High-level resistance | 0
  INI, RAL, Susceptible | 2
  INI, RAL, Potential low-level resistance | 0
  INI, RAL, Low-level resistance | 0
  INI, RAL, Intermediate resistance | 0
  INI, RAL, High-level resistance | 0
  NNRTI, DLV, Susceptible | 2
  NNRTI, DLV, Potential low-level resistance | 0
  NNRTI, DLV, Low-level resistance | 0
  NNRTI, DLV, Intermediate resistance | 0
  NNRTI, DLV, High-level resistance | 0
  NNRTI, EFV, Susceptible | 0
  NNRTI, EFV, Potential low-level resistance | 0
  NNRTI, EFV, Low-level resistance | 1
  NNRTI, EFV, Intermediate resistance | 0
  NNRTI, EFV, High-level resistance | 1
  NNRTI, ETR, Susceptible | 0
  NNRTI, ETR, Potential low-level resistance | 0
  NNRTI, ETR, Low-level resistance | 1
  NNRTI, ETR, Intermediate resistance | 0
  NNRTI, ETR, High-level resistance | 1
  NNRTI, NVP, Susceptible | 0
  NNRTI, NVP, Potential low-level resistance | 0
  NNRTI, NVP, Low-level resistance | 0
  NNRTI, NVP, Intermediate resistance | 1
  NNRTI, NVP, High-level resistance | 1
  NNRTI, RPV, Susceptible | 0
  NNRTI, RPV, Potential low-level resistance | 0
  NNRTI, RPV, Low-level resistance | 0
  NNRTI, RPV, Intermediate resistance | 1
  NNRTI, RPV, High-level resistance | 1
  NRTI, 3TC, Susceptible | 2
  NRTI, 3TC, Potential low-level resistance | 0
  NRTI, 3TC, Low-level resistance | 0
  NRTI, 3TC, Intermediate resistance | 0
  NRTI, 3TC, High-level resistance | 0
  NRTI, ABC, Susceptible | 2
  NRTI, ABC, Potential low-level resistance | 0
  NRTI, ABC, Low-level resistance | 0
  NRTI, ABC, Intermediate resistance | 0
  NRTI, ABC, High-level resistance | 0
  NRTI, FTC, Susceptible | 2
  NRTI, FTC, Potential low-level resistance | 0
  NRTI, FTC, Low-level resistance | 0
  NRTI, FTC, Intermediate resistance | 0
  NRTI, FTC, High-level resistance | 0
  NRTI, TDF, Susceptible | 2
  NRTI, TDF, Potential low-level resistance | 0
  NRTI, TDF, Low-level resistance | 0
  NRTI, TDF, Intermediate resistance | 0
  NRTI, TDF, High-level resistance | 0
  NRTI, ZDV, Susceptible | 2
  NRTI, ZDV, Potential low-level resistance | 0
  NRTI, ZDV, Low-level resistance | 0
  NRTI, ZDV, Intermediate resistance | 0
  NRTI, ZDV, High-level resistance | 0
  NRTI, d4T, Susceptible | 2
  NRTI, d4T, Potential low-level resistance | 0
  NRTI, d4T, Low-level resistance | 0
  NRTI, d4T, Intermediate resistance | 0
  NRTI, d4T, High-level resistance | 0
  NRTI, ddI, Susceptible | 2
  NRTI, ddI, Potential low-level resistance | 0
  NRTI, ddI, Low-level resistance | 0
  NRTI, ddI, Intermediate resistance | 0
  NRTI, ddI, High-level resistance | 0
  PI, ATV/r, Susceptible | 2
  PI, ATV/r, Potential low-level resistance | 0
  PI, ATV/r, Low-level resistance | 0
  PI, ATV/r, Intermediate resistance | 0
  PI, ATV/r, High-level resistance | 0
  PI, DRV/r, Susceptible | 2
  PI, DRV/r, Potential low-level resistance | 0
  PI, DRV/r, Low-level resistance | 0
  PI, DRV/r, Intermediate resistance | 0
  PI, DRV/r, High-level resistance | 0
  PI, FPV/r, Susceptible | 2
  PI, FPV/r, Potential low-level resistance | 0
  PI, FPV/r, Low-level resistance | 0
  PI, FPV/r, Intermediate resistance | 0
  PI, FPV/r, High-level resistance | 0
  PI, IDV/r, Susceptible | 2
  PI, IDV/r, Potential low-level resistance | 0
  PI, IDV/r, Low-level resistance | 0
  PI, IDV/r, Intermediate resistance | 0
  PI, IDV/r, High-level resistance | 0
  PI, LPV/r, Susceptible | 2
  PI, LPV/r, Potential low-level resistance | 0
  PI, LPV/r, Low-level resistance | 0
  PI, LPV/r, Intermediate resistance | 0
  PI, LPV/r, High-level resistance | 0
  PI, NFV, Susceptible | 2
  PI, NFV, Potential low-level resistance | 0
  PI, NFV, Low-level resistance | 0
  PI, NFV, Intermediate resistance | 0
  PI, NFV, High-level resistance | 0
  PI, RTV, Susceptible | 2
  PI, RTV, Potential low-level resistance | 0
  PI, RTV, Low-level resistance | 0
  PI, RTV, Intermediate resistance | 0
  PI, RTV, High-level resistance | 0
  PI, SQV/r, Susceptible | 2
  PI, SQV/r, Potential low-level resistance | 0
  PI, SQV/r, Low-level resistance | 0
  PI, SQV/r, Intermediate resistance | 0
  PI, SQV/r, High-level resistance | 0
  PI, TPV/r, Susceptible | 2
  PI, TPV/r, Potential low-level resistance | 0
  PI, TPV/r, Low-level resistance | 0
  PI, TPV/r, Intermediate resistance | 0
  PI, TPV/r, High-level resistance | 0

22. Secondary Outcome: Number of Participants With Genotypic Resistance-CAR Arm Through Late Switch Phase
Description: Plasma samples were collected for drug resistance testing. Genotypic Resistance data for the following drugs (DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r, TPV/r) in participants Meeting CVW Criteria has been presented.
Time Frame: Post-Late switch (LS) Baseline (Week 52) up to Week 148
Population: The analysis was performed on the Late Switch (LS) CVW resistance Population which was comprised of all participants in the LS ITT-E Population who met CVW through the end of visit window (Week 48, Week 100 or Week 148) and had available on-treatment genotypic resistance data at the time CVW criterion is met. Only those participants with data available at the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1
Participants
  INI, DTG, Susceptible | 1
  INI, DTG, Potential low-level resistance | 0
  INI, DTG, Low-level resistance | 0
  INI, DTG, Intermediate resistance | 0
  INI, DTG, High-level resistance | 0
  INI, EVG, Susceptible | 1
  INI, EVG, Potential low-level resistance | 0
  INI, EVG, Low-level resistance | 0
  INI, EVG, Intermediate resistance | 0
  INI, EVG, High-level resistance | 0
  INI, RAL, Susceptible | 1
  INI, RAL, Potential low-level resistance | 0
  INI, RAL, Low-level resistance | 0
  INI, RAL, Intermediate resistance | 0
  INI, RAL, High-level resistance | 0
  NNRTI, DLV, Susceptible | 1
  NNRTI, DLV, Potential low-level resistance | 0
  NNRTI, DLV, Low-level resistance | 0
  NNRTI, DLV, Intermediate resistance | 0
  NNRTI, DLV, High-level resistance | 0
  NNRTI, EFV, Susceptible | 0
  NNRTI, EFV, Potential low-level resistance | 0
  NNRTI, EFV, Low-level resistance | 0
  NNRTI, EFV, Intermediate resistance | 0
  NNRTI, EFV, High-level resistance | 1
  NNRTI, ETR, Susceptible | 0
  NNRTI, ETR, Potential low-level resistance | 0
  NNRTI, ETR, Low-level resistance | 0
  NNRTI, ETR, Intermediate resistance | 1
  NNRTI, ETR, High-level resistance | 0
  NNRTI, NVP, Susceptible | 0
  NNRTI, NVP, Potential low-level resistance | 0
  NNRTI, NVP, Low-level resistance | 0
  NNRTI, NVP, Intermediate resistance | 0
  NNRTI, NVP, High-level resistance | 1
  NNRTI, RPV, Susceptible | 0
  NNRTI, RPV, Potential low-level resistance | 0
  NNRTI, RPV, Low-level resistance | 0
  NNRTI, RPV, Intermediate resistance | 0
  NNRTI, RPV, High-level resistance | 1
  NRTI, 3TC, Susceptible | 1
  NRTI, 3TC, Potential low-level resistance | 0
  NRTI, 3TC, Low-level resistance | 0
  NRTI, 3TC, Intermediate resistance | 0
  NRTI, 3TC, High-level resistance | 0
  NRTI, ABC, Susceptible | 1
  NRTI, ABC, Potential low-level resistance | 0
  NRTI, ABC, Low-level resistance | 0
  NRTI, ABC, Intermediate resistance | 0
  NRTI, ABC, High-level resistance | 0
  NRTI, FTC, Susceptible | 1
  NRTI, FTC, Potential low-level resistance | 0
  NRTI, FTC, Low-level resistance | 0
  NRTI, FTC, Intermediate resistance | 0
  NRTI, FTC, High-level resistance | 0
  NRTI, TDF, Susceptible | 1
  NRTI, TDF, Potential low-level resistance | 0
  NRTI, TDF, Low-level resistance | 0
  NRTI, TDF, Intermediate resistance | 0
  NRTI, TDF, High-level resistance | 0
  NRTI, ZDV, Susceptible | 1
  NRTI, ZDV, Potential low-level resistance | 0
  NRTI, ZDV, Low-level resistance | 0
  NRTI, ZDV, Intermediate resistance | 0
  NRTI, ZDV, High-level resistance | 0
  NRTI, d4T, Susceptible | 1
  NRTI, d4T, Potential low-level resistance | 0
  NRTI, d4T, Low-level resistance | 0
  NRTI, d4T, Intermediate resistance | 0
  NRTI, d4T, High-level resistance | 0
  NRTI, ddI, Susceptible | 1
  NRTI, ddI, Potential low-level resistance | 0
  NRTI, ddI, Low-level resistance | 0
  NRTI, ddI, Intermediate resistance | 0
  NRTI, ddI, High-level resistance | 0
  PI, ATV/r, Susceptible | 1
  PI, ATV/r, Potential low-level resistance | 0
  PI, ATV/r, Low-level resistance | 0
  PI, ATV/r, Intermediate resistance | 0
  PI, ATV/r, High-level resistance | 0
  PI, DRV/r, Susceptible | 1
  PI, DRV/r, Potential low-level resistance | 0
  PI, DRV/r, Low-level resistance | 0
  PI, DRV/r, Intermediate resistance | 0
  PI, DRV/r, High-level resistance | 0
  PI, FPV/r, Susceptible | 1
  PI, FPV/r, Potential low-level resistance | 0
  PI, FPV/r, Low-level resistance | 0
  PI, FPV/r, Intermediate resistance | 0
  PI, FPV/r, High-level resistance | 0
  PI, IDV/r, Susceptible | 1
  PI, IDV/r, Potential low-level resistance | 0
  PI, IDV/r, Low-level resistance | 0
  PI, IDV/r, Intermediate resistance | 0
  PI, IDV/r, High-level resistance | 0
  PI, LPV/r, Susceptible | 1
  PI, LPV/r, Potential low-level resistance | 0
  PI, LPV/r, Low-level resistance | 0
  PI, LPV/r, Intermediate resistance | 0
  PI, LPV/r, High-level resistance | 0
  PI, NFV, Susceptible | 1
  PI, NFV, Potential low-level resistance | 0
  PI, NFV, Low-level resistance | 0
  PI, NFV, Intermediate resistance | 0
  PI, NFV, High-level resistance | 0
  PI, RTV, Susceptible | 1
  PI, RTV, Potential low-level resistance | 0
  PI, RTV, Low-level resistance | 0
  PI, RTV, Intermediate resistance | 0
  PI, RTV, High-level resistance | 0
  PI, SQV/r, Susceptible | 1
  PI, SQV/r, Potential low-level resistance | 0
  PI, SQV/r, Low-level resistance | 0
  PI, SQV/r, Intermediate resistance | 0
  PI, SQV/r, High-level resistance | 0
  PI, TPV/r, Susceptible | 1
  PI, TPV/r, Potential low-level resistance | 0
  PI, TPV/r, Low-level resistance | 0
  PI, TPV/r, Intermediate resistance | 0
  PI, TPV/r, High-level resistance | 0

23. Secondary Outcome: Number of Participants With Phenotypic Resistance-Early Switch Phase
Description: Plasma samples were collected for drug resistance testing. Phenotypic Resistance data for the following drugs (DTG, RAL, EVG, RPV, ETR, 3TC, ABC, FTC, TDF, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, SQV/r, TPV/r) in participants Meeting CVW criteria has been presented.
Time Frame: Up to Week 52
Population: The analysis was performed on the CVW resistance Population which was comprised of all participants in the ITT-E Population who met CVW through the end of visit window (Week 48, Week 100 or Week 148) and have available on-treatment genotypic resistance data at the time CVW criterion is met. Only participants from the DTG + RPV were analyzed as the CAR participants did not receive study treatment until Week 52.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1 | 0
Participants
  NNRTI, RPV, Resistant | 0 |
  NNRTI, RPV, Sensitive | 1 |
  NNRTI, ETR, Resistant | 0 |
  NNRTI, ETR, Partially Sensitive | 0 |
  NNRTI, ETR, Sensitive | 1 |
  NNRTI, DLV, Resistant | 0 |
  NNRTI, DLV, Sensitive | 1 |
  NNRTI, EFV, Resistant | 0 |
  NNRTI, EFV, Sensitive | 1 |
  NNRTI, NVP, Resistant | 0 |
  NNRTI, NVP, Sensitive | 1 |
  NRTI, 3TC, Resistant | 0 |
  NRTI, 3TC, Sensitive | 1 |
  NRTI, ABC, Resistant | 0 |
  NRTI, ABC, Partially Sensitive | 0 |
  NRTI, ABC, Sensitive | 1 |
  NRTI, TDF, Resistant | 0 |
  NRTI, TDF, Partially Sensitive | 0 |
  NRTI, TDF, Sensitive | 1 |
  NRTI, d4T, Resistant | 0 |
  NRTI, d4T, Sensitive | 1 |
  NRTI, ddI, Resistant | 0 |
  NRTI, ddI, Partially Sensitive | 0 |
  NRTI, ddI, Sensitive | 1 |
  NRTI, FTC, Resistant | 0 |
  NRTI, FTC, Sensitive | 1 |
  NRTI, ZDV, Resistant | 0 |
  NRTI, ZDV, Sensitive | 1 |
  PI, ATV/r, Resistant | 0 |
  PI, ATV/r, Sensitive | 1 |
  PI, DRV/r, Resistant | 0 |
  PI, DRV/r, Partially Sensitive | 0 |
  PI, DRV/r, Sensitive | 1 |
  PI, FPV/r, Resistant | 0 |
  PI, FPV/r, Partially Sensitive | 0 |
  PI, FPV/r, Sensitive | 1 |
  PI, IDV/r, Resistant | 0 |
  PI, IDV/r, Sensitive | 1 |
  PI, LPV/r, Resistant | 0 |
  PI, LPV/r, Partially Sensitive | 0 |
  PI, LPV/r, Sensitive | 1 |
  PI, SQV/r, Resistant | 0 |
  PI, SQV/r, Partially Sensitive | 0 |
  PI, SQV/r, Sensitive | 1 |
  PI, TPV/r, Resistant | 0 |
  PI, TPV/r, Partially Sensitive | 0 |
  PI, TPV/r, Sensitive | 1 |
  PI, NFV, Resistant | 0 |
  PI, NFV, Sensitive | 1 |
  PI, RTV, Resistant | 0 |
  PI, RTV, Sensitive | 1 |

24. Secondary Outcome: Number of Participants With Phenotypic Resistance-DTG+RPV Group Through Early and Late Switch Phase
Description: Plasma samples were collected for drug resistance testing. Phenotypic Resistance data for the following drugs (DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r, TPV/r) in participants Meeting CVW criteria has been presented.
Time Frame: Up to Week 148
Population: CVW resistance Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 2
Participants
  INI, DTG, Resistant: number analyzed (Participants) | 1
  INI, DTG, Resistant | 0
  INI, DTG, Partially Sensitive: number analyzed (Participants) | 1
  INI, DTG, Partially Sensitive | 0
  INI, DTG, Sensitive: number analyzed (Participants) | 1
  INI, DTG, Sensitive | 1
  INI, EVG, Resistant: number analyzed (Participants) | 1
  INI, EVG, Resistant | 0
  INI, EVG, Partially sensitive: number analyzed (Participants) | 1
  INI, EVG, Partially sensitive | 0
  INI, EVG, Sensitive: number analyzed (Participants) | 1
  INI, EVG, Sensitive | 1
  INI, RAL, Resistant: number analyzed (Participants) | 1
  INI, RAL, Resistant | 1
  INI, RAL, Partially sensitive: number analyzed (Participants) | 1
  INI, RAL, Partially sensitive | 0
  INI, RAL, Sensitive: number analyzed (Participants) | 1
  INI, RAL, Sensitive | 0
  NNRTI, DLV, Resistant | 1
  NNRTI, DLV, Partially Sensitive | 0
  NNRTI, DLV, Sensitive | 1
  NNRTI, EFV, Resistant | 1
  NNRTI, EFV, Partially sensitive | 0
  NNRTI, EFV, Sensitive | 1
  NNRTI, ETR, Resistant | 1
  NNRTI, ETR, Partially sensitive | 0
  NNRTI, ETR, Sensitive | 1
  NNRTI, NVP, Resistant | 1
  NNRTI, NVP, Partially sensitive | 0
  NNRTI, NVP, Sensitive | 1
  NNRTI, RPV, Resistant | 1
  NNRTI, RPV, Partially sensitive | 0
  NNRTI, RPV, Sensitive | 1
  NRTI, 3TC, Resistant | 0
  NRTI, 3TC, Partially sensitive | 0
  NRTI, 3TC, Sensitive | 2
  NRTI, ABC, Resistant | 0
  NRTI, ABC, Partially sensitive | 0
  NRTI, ABC, Sensitive | 2
  NRTI, FTC, Resistant | 0
  NRTI, FTC, Partially sensitive | 0
  NRTI, FTC, Sensitive | 2
  NRTI, TDF, Resistant | 0
  NRTI, TDF, Partially sensitive | 0
  NRTI, TDF, Sensitive | 2
  NRTI, ZDV, Resistant | 0
  NRTI, ZDV, Partially sensitive | 0
  NRTI, ZDV, Sensitive | 2
  NRTI, d4T, Resistant | 0
  NRTI, d4T, Partially sensitive | 0
  NRTI, d4T, Sensitive | 2
  NRTI, ddI, Resistant | 0
  NRTI, ddI, Partially sensitive | 0
  NRTI, ddI, Sensitive | 2
  PI, ATV/r, Resistant | 0
  PI, ATV/r, Partially sensitive | 0
  PI, ATV/r, Sensitive | 2
  PI, DRV/r, Resistant | 0
  PI, DRV/r, Partially sensitive | 0
  PI, DRV/r, Sensitive | 2
  PI, FPV/r, Resistant | 0
  PI, FPV/r, Partially sensitive | 0
  PI, FPV/r, Sensitive | 2
  PI, IDV/r, Resistant | 0
  PI, IDV/r, Partially sensitive | 0
  PI, IDV/r, Sensitive | 2
  PI, LPV/r, Resistant | 0
  PI, LPV/r, Partially sensitive | 0
  PI, LPV/r, Sensitive | 2
  PI, NFV, Resistant | 0
  PI, NFV, Partially sensitive | 0
  PI, NFV, Sensitive | 2
  PI, RTV, Resistant | 0
  PI, RTV, Partially sensitive | 0
  PI, RTV, Sensitive | 2
  PI, SQV/r, Resistant | 0
  PI, SQV/r, Partially sensitive | 0
  PI, SQV/r, Sensitive | 2
  PI, TPV/r, Resistant | 0
  PI, TPV/r, Partially sensitive | 0
  PI, TPV/r, Sensitive | 2

25. Secondary Outcome: Number of Participants With Phenotypic Resistance-CAR Group Through Late Switch Phase
Description: as for outcome 24
Time Frame: Post-LS Baseline (Week 52) up to Week 148
Population: LS CVW resistance Population
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1
Participants
  NNRTI, DLV, Resistant | 1
  NNRTI, DLV, Partially Sensitive | 0
  NNRTI, DLV, Sensitive | 0
  NNRTI, EFV, Resistant | 1
  NNRTI, EFV, Partially sensitive | 0
  NNRTI, EFV, Sensitive | 0
  NNRTI, ETR, Resistant | 0
  NNRTI, ETR, Partially sensitive | 1
  NNRTI, ETR, Sensitive | 0
  NNRTI, NVP, Resistant | 1
  NNRTI, NVP, Partially sensitive | 0
  NNRTI, NVP, Sensitive | 0
  NNRTI, RPV, Resistant | 1
  NNRTI, RPV, Partially sensitive | 0
  NNRTI, RPV, Sensitive | 0
  NRTI, 3TC, Resistant | 0
  NRTI, 3TC, Partially sensitive | 0
  NRTI, 3TC, Sensitive | 1
  NRTI, ABC, Resistant | 0
  NRTI, ABC, Partially sensitive | 0
  NRTI, ABC, Sensitive | 1
  NRTI, FTC, Resistant | 0
  NRTI, FTC, Partially sensitive | 0
  NRTI, FTC, Sensitive | 1
  NRTI, TDF, Resistant | 0
  NRTI, TDF, Partially sensitive | 0
  NRTI, TDF, Sensitive | 1
  NRTI, ZDV, Resistant | 0
  NRTI, ZDV, Partially sensitive | 0
  NRTI, ZDV, Sensitive | 1
  NRTI, d4T, Resistant | 0
  NRTI, d4T, Partially sensitive | 0
  NRTI, d4T, Sensitive | 1
  NRTI, ddI, Resistant | 0
  NRTI, ddI, Partially sensitive | 0
  NRTI, ddI, Sensitive | 1
  PI, ATV/r, Resistant | 0
  PI, ATV/r, Partially sensitive | 0
  PI, ATV/r, Sensitive | 1
  PI, DRV/r, Resistant | 0
  PI, DRV/r, Partially sensitive | 0
  PI, DRV/r, Sensitive | 1
  PI, FPV/r, Resistant | 0
  PI, FPV/r, Partially sensitive | 0
  PI, FPV/r, Sensitive | 1
  PI, IDV/r, Resistant | 0
  PI, IDV/r, Partially sensitive | 0
  PI, IDV/r, Sensitive | 1
  PI, LPV/r, Resistant | 0
  PI, LPV/r, Partially sensitive | 0
  PI, LPV/r, Sensitive | 1
  PI, NFV, Resistant | 0
  PI, NFV, Partially sensitive | 0
  PI, NFV, Sensitive | 1
  PI, RTV, Resistant | 0
  PI, RTV, Partially sensitive | 0
  PI, RTV, Sensitive | 1
  PI, SQV/r, Resistant | 0
  PI, SQV/r, Partially sensitive | 0
  PI, SQV/r, Sensitive | 1
  PI, TPV/r, Resistant | 0
  PI, TPV/r, Partially sensitive | 0
  PI, TPV/r, Sensitive | 1

26. Secondary Outcome: Pre-dose Concentrations of DTG and RPV in Participants Switching to DTG + RPV - DTG+RPV Group Through Early and Late Switch Phase
Description: Two separate blood samples for DTG and RPV were collected pre-dose at Weeks 4, 24, 48, 56, 76 and 100. Pre-dose concentrations of DTG and RPV at Weeks 4, 24, 48, 56, 76 and 100 is summarized for the participants switching to DTG + RPV in the early+late switch phase.
Time Frame: Pre-dose at Week 4, 24, 48, 56, 76 and 100
Population: The analysis was performed on the Pharmacokinetic (PK) Parameter Population which consisted of all participants who received DTG +RPV and provided at least one evaluable estimate of predose concentration (C0). Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: ug/ L
Groups:
- DTG 50 mg: Participants received DTG 50 mg + RPV 25 mg together once daily, with a meal, in an open-label fashion up to Week 148 during early switch and late switch phase.
- RPV 25 mg: Participants received DTG 50 mg +RPV 25 mg together once daily, with a meal, in an open-label fashion up to Week 148 during early switch and late switch phase.
Arm/Group | DTG 50 mg | RPV 25 mg
Number analyzed (Participants) | 254 | 254
ug/ L
  Week 4: number analyzed (Participants) | 176 | 175
  Week 4 | 1578.88 (1170.967) | 79.50 (38.230)
  Week 24: number analyzed (Participants) | 207 | 207
  Week 24 | 1447.23 (917.677) | 90.21 (46.302)
  Week 48: number analyzed (Participants) | 215 | 215
  Week 48 | 1384.36 (889.829) | 91.41 (47.073)
  Week 56: number analyzed (Participants) | 214 | 213
  Week 56 | 1637.74 (1063.391) | 90.55 (45.686)
  Week 76: number analyzed (Participants) | 219 | 219
  Week 76 | 1507.81 (913.263) | 92.51 (46.223)
  Week 100: number analyzed (Participants) | 220 | 221
  Week 100 | 1532.10 (916.975) | 91.98 (44.683)

27. Secondary Outcome: Pre-dose Concentrations of DTG and RPV in Participants Switching to DTG + RPV - CAR Group Through Late Switch Phase
Description: Two separate blood samples for DTG and RPV were collected pre-dose at Weeks 56, 76 and 100. Pre-dose concentrations of DTG and RPV at Weeks 56, 76 and 100 is summarized for the participants switching to DTG + RPV in the late switch phase.
Time Frame: Pre-dose at Weeks 56, 76 and 100
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ug/ L
Groups:
- CAR-DTG 50 mg: Participants from CAR arm received DTG 50 mg + RPV 25 mg together once daily, with a meal, in an open-label fashion from Week 52 to Week 148 during late switch phase.
- CAR-RPV 25 mg: Participants from CAR arm received DTG 50 mg +RPV 25 mg together once daily, with a meal, in an open-label fashion from Week 52 to Week 148 during late switch phase.
Arm/Group | CAR-DTG 50 mg | CAR-RPV 25 mg
Number analyzed (Participants) | 226 | 226
ug/ L
  Week 56: number analyzed (Participants) | 203 | 203
  Week 56 | 1544.75 (1049.595) | 77.27 (38.931)
  Week 76: number analyzed (Participants) | 210 | 210
  Week 76 | 1806.77 (1019.300) | 91.46 (48.568)
  Week 100: number analyzed (Participants) | 215 | 215
  Week 100 | 1881.97 (1160.587) | 90.89 (47.762)

28. Secondary Outcome: Pre-dose Concentrations of DTG and RPV in the First 20 Participants Who Switch From Efavirenz (EFV) or Nevirapine (NVP) to DTG + RPV
Description: Two blood samples were collected pre-dose for DTG and RPV at Weeks 2 and 8 only for the first 20 participants who switch from EFV or NVP to DTG+RPV, in addition to the pre-dose blood sample collected at Week 4 for all participants. One blood sample was collected pre-dose for EFV or NVP at Week 2 for the first 20 participants who switch from EFV or NVP to DTG + RPV. PK Parameter NNRTI Subset Extra Sampling Population consisted of the first approximately 20 participants in the PK Parameter NNRTI Subset population who have extra PK samples at weeks 2 and 8.
Time Frame: Pre-dose at Weeks 2, 4 and 8
Population: PK Parameter NNRTI Subset extra sampling Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: ug/ L
Groups:
- DTG 50 mg: Participants received DTG 50 mg + RPV 25 mg together once daily, with a meal, in an open-label fashion up to Week 52 during early switch phase.
- RPV 25 mg: Participants received DTG 50 mg +RPV 25 mg together once daily, with a meal, in an open-label fashion up to Week 52 during early switch phase.
Arm/Group | DTG 50 mg | RPV 25 mg
Number analyzed (Participants) | 28 | 28
ug/ L
  Week 2: number analyzed (Participants) | 19 | 19
  Week 2 | 834.58 (639.622) | 57.342 (29.5436)
  Week 4: number analyzed (Participants) | 22 | 21
  Week 4 | 1218.23 (842.703) | 78.338 (31.4825)
  Week 8: number analyzed (Participants) | 26 | 26
  Week 8 | 1472.50 (818.774) | 79.652 (40.7546)

29. Secondary Outcome: Percentage of Participants With Plasma HIV 1 RNA <50 c/mL at Week 48 Using Snapshot Algorithm by Baseline Third Agent Treatment Class
Description: Percentage of participants with plasma HIV 1 RNA < 50 c/mL at Week 48 using the FDA snapshot algorithm was assessed by Baseline third agent class to assess the impact of Baseline third agent class (INSTI, NNRTI, or PI) on efficacy, safety and tolerability of DTG +RPV compared to continuation of CAR. Plasma samples were collected for HIV-1 RNA at Baseline (Day 1), Week 4, 8, 12, 24, 36 and 48. The analysis was done using Cochran-Mantel Haenszel test stratified by current antiretroviral third-agent class.
Time Frame: At Week 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Percentage of participants
  NNRTI: number analyzed (Participants) | 144 | 144
  NNRTI | 97 | 93
  INSTI: number analyzed (Participants) | 59 | 49
  INSTI | 92 | 94
  PI: number analyzed (Participants) | 58 | 62
  PI | 91 | 97
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.179, Chi-squared, Corrected — One-sided p-value from weighted least squares chi-squared statistic. A p-value <=0.10 was used to indicate statistically significant evidence of heterogeneity in the difference in proportions across levels of each analysis strata
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; Risk Difference (RD) = 3.5, 95% CI 2-sided [-1.6 to 8.6] — NNRTI: No formal non-inferiority margin has been pre-specified for secondary endpoints
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; Risk Difference (RD) = -2.4, 95% CI 2-sided [-12.1 to 7.4] — INSTI: No formal non-inferiority margin has been pre-specified for secondary endpoints
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; Risk Difference (RD) = -5.4, 95% CI 2-sided [-13.9 to 3.1] — PI: No formal non-inferiority margin has been pre-specified for secondary endpoints

30. Secondary Outcome: Changes From Baseline in CD4+ Lymphocyte Count at Week 48 by Baseline Third Agent Treatment Class
Description: Blood samples were collected and CD4+ cell count assessment by flow cytometry was carried out at Baseline (Day 1) and Week 48 to assess the impact of Baseline third agent class (INSTI, NNRTI, or PI) on efficacy, safety and tolerability of DTG +RPV compared to continuation of CAR. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per mm^3
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Cells per mm^3
  NNRTI: number analyzed (Participants) | 139 | 133
  NNRTI | 49.7 (166.40) | 24.3 (160.32)
  INSTI: number analyzed (Participants) | 53 | 46
  INSTI | -11.2 (176.56) | 10.3 (155.53)
  PI: number analyzed (Participants) | 53 | 61
  PI | 10.5 (163.67) | 12.2 (163.32)

31. Secondary Outcome: Number of Participants With Any AE, AELD or AE With Grade 1, 2, 3 or 4 Toxicity Over 48 Weeks by Baseline Third Agent Treatment Class
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with any AE, AELD or AE with maximum grade toxicity experienced by any one participant over 48 weeks by Baseline third agent class (INSTI, NNRTI, or PI) is summarized. AEs were graded using the Division of AIDS grading. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening.
Time Frame: Up to 48 weeks
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Participants
  Any AE, NNRTI: number analyzed (Participants) | 144 | 144
  Any AE, NNRTI | 106 | 96
  Any AE, INSTI: number analyzed (Participants) | 59 | 49
  Any AE, INSTI | 47 | 36
  Any AE, PI: number analyzed (Participants) | 58 | 62
  Any AE, PI | 42 | 42
  NNRTI, Maximum toxicity Grade 1 AE: number analyzed (Participants) | 144 | 144
  NNRTI, Maximum toxicity Grade 1 AE | 68 | 76
  NNRTI, Maximum toxicity Grade 2 AE: number analyzed (Participants) | 144 | 144
  NNRTI, Maximum toxicity Grade 2 AE | 30 | 19
  NNRTI, Maximum toxicity Grade 3 AE: number analyzed (Participants) | 144 | 144
  NNRTI, Maximum toxicity Grade 3 AE | 8 | 0
  NNRTI, Maximum toxicity Grade 4 AE: number analyzed (Participants) | 144 | 144
  NNRTI, Maximum toxicity Grade 4 AE | 0 | 1
  INSTI, Maximum toxicity Grade 1 AE: number analyzed (Participants) | 59 | 49
  INSTI, Maximum toxicity Grade 1 AE | 27 | 20
  INSTI, Maximum toxicity Grade 2 AE: number analyzed (Participants) | 59 | 49
  INSTI, Maximum toxicity Grade 2 AE | 15 | 15
  INSTI, Maximum toxicity Grade 3 AE: number analyzed (Participants) | 59 | 49
  INSTI, Maximum toxicity Grade 3 AE | 5 | 1
  INSTI, Maximum toxicity Grade 4 AE: number analyzed (Participants) | 59 | 49
  INSTI, Maximum toxicity Grade 4 AE | 0 | 0
  PI, Maximum toxicity Grade 1 AE: number analyzed (Participants) | 58 | 62
  PI, Maximum toxicity Grade 1 AE | 24 | 26
  PI, Maximum toxicity Grade 2 AE: number analyzed (Participants) | 58 | 62
  PI, Maximum toxicity Grade 2 AE | 14 | 13
  PI, Maximum toxicity Grade 3 AE: number analyzed (Participants) | 58 | 62
  PI, Maximum toxicity Grade 3 AE | 3 | 3
  PI, Maximum toxicity Grade 4 AE: number analyzed (Participants) | 58 | 62
  PI, Maximum toxicity Grade 4 AE | 1 | 0
  AELD, NNRTI: number analyzed (Participants) | 144 | 144
  AELD, NNRTI | 5 | 1
  AELD, INSTI: number analyzed (Participants) | 59 | 49
  AELD, INSTI | 4 | 0
  AELD, PI: number analyzed (Participants) | 58 | 62
  AELD, PI | 3 | 0

32. Secondary Outcome: Number of Participants With Maximum Post-baseline Emergent Chemistry Toxicities Over 48 Weeks by Baseline Third Agent Treatment Class
Description: Blood samples were collected at Baseline (Day 1) and at Weeks 4, 8, 12, 24, 36 and 48 to evaluate ALT, albumin, ALP, AST, total bilirubin, chloride, creatinine, glucose, potassium, phosphate, sodium, BUN, total carbon dioxide, lipase, creatine phosphokinase and creatinine clearance. Number of participants who experienced maximum toxicity grade post-baseline in chemistry parameters over 48 weeks by Baseline third agent treatment class (INSTI, NNRTI, PI) is summarized. Clinical chemistry toxicities were graded using the DAIDS grading. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening.
Time Frame: Up to 48 weeks
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Participants
  NNRTI, Grade 1: number analyzed (Participants) | 144 | 144
  NNRTI, Grade 1 | 51 | 52
  NNRTI, Grade 2: number analyzed (Participants) | 144 | 144
  NNRTI, Grade 2 | 31 | 40
  NNRTI, Grade 3: number analyzed (Participants) | 144 | 144
  NNRTI, Grade 3 | 7 | 4
  NNRTI, Grade 4: number analyzed (Participants) | 144 | 144
  NNRTI, Grade 4 | 1 | 5
  INSTI, Grade 1: number analyzed (Participants) | 59 | 49
  INSTI, Grade 1 | 19 | 11
  INSTI, Grade 2: number analyzed (Participants) | 59 | 49
  INSTI, Grade 2 | 23 | 18
  INSTI, Grade 3: number analyzed (Participants) | 59 | 49
  INSTI, Grade 3 | 3 | 3
  INSTI, Grade 4: number analyzed (Participants) | 59 | 49
  INSTI, Grade 4 | 0 | 2
  PI, Grade 1: number analyzed (Participants) | 58 | 62
  PI, Grade 1 | 22 | 17
  PI, Grade 2: number analyzed (Participants) | 58 | 62
  PI, Grade 2 | 18 | 21
  PI, Grade 3: number analyzed (Participants) | 58 | 62
  PI, Grade 3 | 1 | 9
  PI, Grade 4: number analyzed (Participants) | 58 | 62
  PI, Grade 4 | 0 | 3

33. Secondary Outcome: Number of Participants With Maximum Post-baseline Emergent Hematology Toxicities Over 48 Weeks by Baseline Third Agent Treatment Class
Description: Blood samples were collected at Baseline (Day 1) and at Weeks 4, 8, 12, 24, 36 and 48 to evaluate hemoglobin, hematocrit, basophils, eosinophils, lymphocytes, monocytes, neutrophils, MCV, RBC count, WBC count and platelet count. Number of participants who experienced maximum toxicity grade post-baseline in hematology parameters over 48 weeks by Baseline third agent treatment class (INSTI, NNRTI, PI) was summarized. Hematology toxicities were graded using the DAIDS grading. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening.
Time Frame: Up to 48 weeks
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Participants
  NNRTI; Grade 1: number analyzed (Participants) | 144 | 144
  NNRTI; Grade 1 | 7 | 6
  NNRTI; Grade 2: number analyzed (Participants) | 144 | 144
  NNRTI; Grade 2 | 1 | 2
  NNRTI; Grade 3: number analyzed (Participants) | 144 | 144
  NNRTI; Grade 3 | 1 | 0
  NNRTI; Grade 4: number analyzed (Participants) | 144 | 144
  NNRTI; Grade 4 | 1 | 0
  INI; Grade 1: number analyzed (Participants) | 59 | 49
  INI; Grade 1 | 1 | 1
  INI; Grade 2: number analyzed (Participants) | 59 | 49
  INI; Grade 2 | 0 | 0
  INI; Grade 3: number analyzed (Participants) | 59 | 49
  INI; Grade 3 | 0 | 0
  INI; Grade 4: number analyzed (Participants) | 59 | 49
  INI; Grade 4 | 0 | 0
  PI; Grade 1: number analyzed (Participants) | 58 | 62
  PI; Grade 1 | 3 | 4
  PI; Grade 2: number analyzed (Participants) | 58 | 62
  PI; Grade 2 | 1 | 0
  PI; Grade 3: number analyzed (Participants) | 58 | 62
  PI; Grade 3 | 2 | 0
  PI; Grade 4: number analyzed (Participants) | 58 | 62
  PI; Grade 4 | 0 | 0

34. Secondary Outcome: Number of Participants With Observed Genotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class
Description: For all participants who meet virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were to be analyzed in an attempt to obtain genotype data on as many samples as possible. Samples for drug resistance testing (genotypic) were to be collected at Day 1. Number of participants with genotypic resistance to CAR and to DTG or RPV for those meeting virologic withdrawal criteria in subgroups stratified based on Baseline third agent treatment class (INSTI, NNRTI, PI) were to be summarized.
Time Frame: Week 48
Population: CVW resistance Population. This outcome has not been analyzed as the number of participants was low (1 CVW per arm) and summaries by Baseline third agent were not provided. Therefore, data are not available for this outcome measure due to the insufficient number of participants with events.
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Number of Participants With Observed Phenotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class
Description: For all participants who meet virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were to be analyzed in an attempt to obtain phenotype data on as many samples as possible. Samples for drug resistance testing (phenotypic) were to be collected at Day 1. Number of participants with phenotypic resistance to CAR and to DTG or RPV for those meeting virologic withdrawal criteria in subgroups stratified based on Baseline third agent treatment class (INSTI, NNRTI, PI) were to be summarized.
Time Frame: Week 48
Population: CVW resistance Population. This outcome was not analyzed as the number of participants was low (1 CVW per arm) and summaries by Baseline third agent were not provided. Therefore, data are not available for this outcome measure due to the insufficient number of participants with events.
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Change From Baseline in Fasting Lipids at Weeks 24 and 48 by Baseline Third Agent Treatment Class
Description: Blood samples were collected at Baseline (Day 1), Weeks 24 and 48 to assess fasting lipids which included total cholesterol (CHO), LDL cholesterol, HDL cholesterol and triglycerides. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Weeks 24 and 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
mmol/L
  CHO, Week 24, overall: number analyzed (Participants) | 237 | 229
  CHO, Week 24, overall | 1.015 (15.7472) | 1.300 (12.2269)
  CHO, Week 48, overall: number analyzed (Participants) | 237 | 230
  CHO, Week 48, overall | -0.165 (15.9301) | 0.194 (13.1071)
  CHO, Week 24, NNRTI: number analyzed (Participants) | 0 | 132
  CHO, Week 24, NNRTI |  | 1.238 (12.4889)
  CHO, Week 48, NNRTI: number analyzed (Participants) | 0 | 128
  CHO, Week 48, NNRTI |  | 0.281 (12.2469)
  CHO, Week 24, INSTI: number analyzed (Participants) | 0 | 42
  CHO, Week 24, INSTI |  | 1.973 (12.1365)
  CHO, Week 48, INSTI: number analyzed (Participants) | 0 | 44
  CHO, Week 48, INSTI |  | 2.798 (16.1468)
  CHO, Week 24, PI: number analyzed (Participants) | 0 | 55
  CHO, Week 24, PI |  | 0.936 (11.8530)
  CHO, Week 48, PI: number analyzed (Participants) | 0 | 58
  CHO, Week 48, PI |  | -1.971 (12.2195)
  HDL CHO direct, Overall, Week 24: number analyzed (Participants) | 237 | 229
  HDL CHO direct, Overall, Week 24 | 0.557 (19.4929) | -2.533 (16.3641)
  HDL CHO direct, Overall, Week 48: number analyzed (Participants) | 237 | 230
  HDL CHO direct, Overall, Week 48 | 6.384 (20.9244) | 4.723 (18.3253)
  HDL CHO direct, NNRTI, Week 24: number analyzed (Participants) | 0 | 132
  HDL CHO direct, NNRTI, Week 24 |  | -2.562 (15.3521)
  HDL CHO direct, NNRTI, Week 48: number analyzed (Participants) | 0 | 128
  HDL CHO direct, NNRTI, Week 48 |  | 4.307 (17.8013)
  HDL CHO direct, INSTI, Week 24: number analyzed (Participants) | 0 | 42
  HDL CHO direct, INSTI, Week 24 |  | -3.097 (20.0002)
  HDL CHO direct, INSTI, Week 48: number analyzed (Participants) | 0 | 44
  HDL CHO direct, INSTI, Week 48 |  | 5.386 (20.6791)
  HDL CHO direct, PI, Week 24: number analyzed (Participants) | 0 | 55
  HDL CHO direct, PI, Week 24 |  | -2.031 (15.9582)
  HDL CHO direct, PI, Week 48: number analyzed (Participants) | 0 | 58
  HDL CHO direct, PI, Week 48 |  | 5.140 (17.8779)
  LDL CHO calculation, Overall, Week 24: number analyzed (Participants) | 231 | 221
  LDL CHO calculation, Overall, Week 24 | 5.838 (22.9614) | 4.395 (21.6685)
  LDL CHO calculation, Overall, Week 48: number analyzed (Participants) | 229 | 220
  LDL CHO calculation, Overall, Week 48 | 1.137 (23.3849) | -0.598 (20.6931)
  LDL CHO calculation, NNRTI, Week 24: number analyzed (Participants) | 0 | 129
  LDL CHO calculation, NNRTI, Week 24 |  | 5.959 (21.5692)
  LDL CHO calculation, NNRTI, Week 48: number analyzed (Participants) | 0 | 124
  LDL CHO calculation, NNRTI, Week 48 |  | 0.747 (19.2299)
  LDL CHO calculation, INSTI, Week 24: number analyzed (Participants) | 0 | 40
  LDL CHO calculation, INSTI, Week 24 |  | 3.787 (17.6755)
  LDL CHO calculation, INSTI, Week 48: number analyzed (Participants) | 0 | 42
  LDL CHO calculation, INSTI, Week 48 |  | 2.647 (24.0430)
  LDL CHO calculation, PI, Week 24: number analyzed (Participants) | 0 | 52
  LDL CHO calculation, PI, Week 24 |  | 0.983 (24.5052)
  LDL CHO calculation, PI, Week 48: number analyzed (Participants) | 0 | 54
  LDL CHO calculation, PI, Week 48 |  | -6.212 (20.4774)
  Triglycerides, Overall, Week 24: number analyzed (Participants) | 237 | 229
  Triglycerides, Overall, Week 24 | -0.825 (42.5565) | 9.379 (45.5529)
  Triglycerides, Overall, Week 48: number analyzed (Participants) | 237 | 230
  Triglycerides, Overall, Week 48 | 1.169 (51.9844) | 7.183 (44.7044)
  Triglycerides, NNRTI, Week 24: number analyzed (Participants) | 0 | 132
  Triglycerides, NNRTI, Week 24 |  | 4.962 (40.6201)
  Triglycerides, NNRTI, Week 48: number analyzed (Participants) | 0 | 128
  Triglycerides, NNRTI, Week 48 |  | 5.248 (41.7728)
  Triglycerides, INSTI, Week 24: number analyzed (Participants) | 0 | 42
  Triglycerides, INSTI, Week 24 |  | 18.204 (47.2348)
  Triglycerides, INSTI, Week 48: number analyzed (Participants) | 0 | 44
  Triglycerides, INSTI, Week 48 |  | 14.627 (56.2824)
  Triglycerides, PI, Week 24: number analyzed (Participants) | 0 | 55
  Triglycerides, PI, Week 24 |  | 13.241 (54.2327)
  Triglycerides, PI, Week 48: number analyzed (Participants) | 0 | 58
  Triglycerides, PI, Week 48 |  | 5.806 (41.2106)

37. Secondary Outcome: Change From Baseline in Pre-specified Treatment Symptoms Using the Symptom Distress Module at Weeks 4, 24 and 48-Early Switch Phase
Description: The Symptom Distress Module, also called the HIV Symptom Index or Symptoms Impact Questionnaire, is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Symptom count is based on which of the 20 symptoms were present in the participant and is the sum of the number of symptoms present and ranges from 0 (none) to 20 (all). Symptom bother score is based on the score for each symptom present ranging from 1 (it doesn't bother me) to 4 (it bothers me a lot). Symptom bother score is the unweighted sum of the bother item scores for each symptom. The symptom bother score ranges from 0 (minimum bother score) to 80 (maximum bother score). Last observation carried forward (LOCF) was used as primary method of analysis. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Weeks 4, 24 and 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Scores on a scale
  Symptom count, Week 4: number analyzed (Participants) | 224 | 229
  Symptom count, Week 4 | -1.1 (4.11) | -0.8 (4.02)
  Symptom count, Week 24: number analyzed (Participants) | 228 | 232
  Symptom count, Week 24 | -0.7 (4.31) | -0.8 (4.64)
  Symptom count, Week 48: number analyzed (Participants) | 228 | 231
  Symptom count, Week 48 | -0.5 (4.33) | -0.4 (4.82)
  Symptom Bother Score, Week 4: number analyzed (Participants) | 224 | 229
  Symptom Bother Score, Week 4 | -2.8 (7.44) | -1.8 (7.24)
  Symptom Bother Score, Week 24: number analyzed (Participants) | 228 | 232
  Symptom Bother Score, Week 24 | -1.8 (8.40) | -1.7 (8.72)
  Symptom Bother Score, Week 48: number analyzed (Participants) | 228 | 231
  Symptom Bother Score, Week 48 | -1.5 (7.97) | -0.7 (9.30)
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.430, ANCOVA — P-value for interaction between treatment group and Baseline symptom bother score (Week 4)
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.039, ANCOVA — P value assessed the difference between treatment groups (Symptom Bother Score - Week 4); Mean Difference (Final Values) = -1.239, 95% CI 2-sided [-2.414 to -0.064] — Estimates were calculated from an ANCOVA model adjusting for age, Baseline third agent, gender, race and Baseline score
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.542, ANCOVA — P-value for interaction between treatment group and Baseline symptom bother score (Week 24)
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.448, ANCOVA — P value assessed the difference between treatment groups (Symptom Bother Score - Week 24); Mean Difference (Final Values) = -0.528, 95% CI 2-sided [-1.896 to 0.840] — Estimates were calculated from an ANCOVA model adjusting for age, Baseline third agent, gender, race and Baseline score
Statistical Analysis 5: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.402, ANCOVA — P-value for interaction between treatment group and Baseline symptom bother score (Week 48)
Statistical Analysis 6: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.164, ANCOVA — P value assessed the difference between treatment groups (Symptom Bother Score - Week 48); Mean Difference (Final Values) = -1.037, 95% CI 2-sided [-2.501 to 0.426] — Estimates were calculated from an ANCOVA model adjusting for age, Baseline third agent, gender, race and Baseline score

38. Secondary Outcome: Change From Baseline in Pre-specified Treatment Symptoms Using the Symptom Distress Module at Weeks 56, 76, 100 and 148-DTG+RPV Group Through Early and Late Switch Phase
Description: The Symptom Distress Module, also called the HIV Symptom Index or Symptoms Impact Questionnaire, is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Symptom count is based on which of the 20 symptoms were present in the participant and is the sum of the number of symptoms present and ranges from 0 (none) to 20 (all). Symptom bother score is based on the score for each symptom present ranging from 1 (it doesn't bother me) to 4 (it bothers me a lot). Symptom bother score is the unweighted sum of the bother item scores for each symptom. The symptom bother score ranges from 0 (minimum bother score) to 80 (maximum bother score). LOCF was used as primary method of analysis. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Weeks 56, 76, 100 and 148
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG + RPV
Number analyzed (Participants) | 228
Scores on a scale
  Symptom count, Week 56 | -0.8 (4.80)
  Symptom count, Week 76 | -0.6 (4.66)
  Symptom count, Week 100 | -0.5 (5.03)
  Symptom count, Week 148 | -0.7 (4.87)
  Symptom Bother Score, Week 56 | -1.8 (9.23)
  Symptom Bother Score, Week 76 | -1.6 (8.70)
  Symptom Bother Score, Week 100 | -1.4 (9.40)
  Symptom Bother Score, Week 148 | -1.7 (9.54)

39. Secondary Outcome: Change From LS Baseline in Pre-specified Treatment Symptoms Using the Symptom Distress Module at Weeks 56, 76, 100 and 148-CAR Group Through Late Switch Phase
Description: The Symptom Distress Module, also called the HIV Symptom Index or Symptoms Impact Questionnaire, is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Symptom count is based on which of the 20 symptoms were present in the participant and is the sum of the number of symptoms present and ranges from 0 (none) to 20 (all). Symptom bother score is based on the score for each symptom present ranging from 1 (it doesn't bother me) to 4 (it bothers me a lot). Symptom bother score is the unweighted sum of the bother item scores for each symptom. The symptom bother score ranges from 0 (minimum bother score) to 80 (maximum bother score). LOCF was used as primary method of analysis. Change from LS Baseline was calculated as value at indicated time point minus LS Baseline value.
Time Frame: At Weeks 56, 76, 100 and 148
Population: LS ITT-E Population comprised of all participants randomized to CAR who received at least one dose of study treatment at or after the Week 52 Switch visit. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 239
Scores on a scale
  Symptom count, Week 56: number analyzed (Participants) | 216
  Symptom count, Week 56 | -0.9 (4.74)
  Symptom count, Week 76: number analyzed (Participants) | 220
  Symptom count, Week 76 | -0.7 (4.29)
  Symptom count, Week 100: number analyzed (Participants) | 220
  Symptom count, Week 100 | -0.4 (5.04)
  Symptom count, Week 148: number analyzed (Participants) | 220
  Symptom count, Week 148 | -0.6 (4.81)
  Symptom Bother Score, Week 56: number analyzed (Participants) | 216
  Symptom Bother Score, Week 56 | -2.1 (7.56)
  Symptom Bother Score, Week 76: number analyzed (Participants) | 220
  Symptom Bother Score, Week 76 | -1.0 (7.61)
  Symptom Bother Score, Week 100: number analyzed (Participants) | 220
  Symptom Bother Score, Week 100 | -0.8 (8.43)
  Symptom Bother Score, Week 148: number analyzed (Participants) | 220
  Symptom Bother Score, Week 148 | -1.0 (8.54)

40. Secondary Outcome: Change From Baseline Treatment Satisfaction Using the HIV Treatment Satisfaction Questionnaire (HIV TSQ) at Weeks 4, 24 and 48-Early Switch Phase
Description: The HIV TSQ is a 10-item self-reported scale that measures overall satisfaction with treatment and by specific domains e.g., convenience, flexibility. Each item is scored 0 to 6 where a higher score indicates the greater improvement in the past few weeks. These items are summed up to produce a treatment satisfaction total score (0 to 60) and 2 subscales: general satisfaction/clinical and lifestyle/ease subscales (0 to 30). The HIV TSQ was administered as a paper questionnaire. Total score, lifestyle/ease score and General satisfaction/clinical sub-score (CS) have been summarized. LOCF was used as primary method of analysis. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Weeks 4, 24 and 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 261 | 255
Score on a scale
  Total score, Week 4: number analyzed (Participants) | 253 | 250
  Total score, Week 4 | 0.0 [-21 to 23] | 0.0 [-22 to 22]
  Total score, Week 24: number analyzed (Participants) | 257 | 252
  Total score, Week 24 | 0.0 [-27 to 23] | 0.0 [-24 to 24]
  Total score, Week 48: number analyzed (Participants) | 257 | 251
  Total score, Week 48 | 0.0 [-27 to 25] | 0.0 [-50 to 23]
  lifestyle/ease Sub-score, Week 4: number analyzed (Participants) | 252 | 249
  lifestyle/ease Sub-score, Week 4 | 0.0 [-11 to 15] | 0.0 [-11 to 7]
  lifestyle/ease Sub-score, Week 24: number analyzed (Participants) | 257 | 251
  lifestyle/ease Sub-score, Week 24 | 0.0 [-18 to 14] | 0.0 [-17 to 10]
  lifestyle/ease Sub-score, Week 48: number analyzed (Participants) | 257 | 250
  lifestyle/ease Sub-score, Week 48 | 0.0 [-18 to 12] | 0.0 [-21 to 11]
  General Satisfaction/CS, Week 4: number analyzed (Participants) | 253 | 250
  General Satisfaction/CS, Week 4 | 0.0 [-13 to 14] | 0.0 [-17 to 15]
  General Satisfaction/CS, Week 24: number analyzed (Participants) | 257 | 252
  General Satisfaction/CS, Week 24 | 0.0 [-12 to 12] | 0.0 [-15 to 15]
  General Satisfaction/CS, Week 48: number analyzed (Participants) | 257 | 251
  General Satisfaction/CS, Week 48 | 0.0 [-13 to 14] | 0.0 [-29 to 14]
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.037, Wilcoxon rank sum test — P-value assessed the HIVTSQs Total Score difference between treatment groups (Week 4)
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.101, Wilcoxon rank sum test — P-value assessed the HIVTSQs Total Score difference between treatment groups (Week 24)
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.042, Wilcoxon rank sum test — P-value assessed the HIVTSQs Total score difference between treatment groups (Week 48)
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.132, Wilcoxon rank sum test — P-value assessed the HIVTSQs lifestyle/ease sub- score difference between treatment groups (Week 4)
Statistical Analysis 5: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.022, Wilcoxon rank sum test — P-value assessed the HIVTSQs lifestyle/ease sub- score difference between treatment groups (Week 24)
Statistical Analysis 6: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.004, Wilcoxon rank sum test — P-value assessed the HIVTSQs lifestyle/ease sub- score difference between treatment groups (Week 48)
Statistical Analysis 7: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.076, Wilcoxon rank sum test — P-value assessed the HIVTSQs General satisfaction/CS sub- score difference between treatment groups (Week 4)
Statistical Analysis 8: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.073, Wilcoxon rank sum test — P-value assessed the HIVTSQs General satisfaction/CS sub- score difference between treatment groups (Week 24)
Statistical Analysis 9: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.547, Wilcoxon rank sum test — P-value assessed the HIVTSQs General satisfaction/CS sub- score difference between treatment groups (Week 48)

41. Secondary Outcome: Change From Baseline Treatment Satisfaction Using the HIV TSQ at Weeks 56, 76, 100 and 148-DTG+RPV Group Through Early and Late Switch Phase
Description: The HIV TSQ is a 10-item self-reported scale that measures overall satisfaction with treatment and by specific domains e.g., convenience, flexibility. Each item is scored 0 (very dissatisfied, inconvenient) to 6 (very satisfied, convenient). The items are summed up to produce a treatment satisfaction total score (0 to 60) and 2 subscale scores: general satisfaction/clinical and lifestyle/ease subscales (0 to 30). Higher scores indicated greater treatment satisfaction as compared to the past few weeks. The HIV TSQ was administered as a paper questionnaire. Change from Baseline is calculated as the value at specified time point minus Baseline value. Total score, lifestyle/ease score and General satisfaction/clinical sub-score (CS) have been summarized. LOCF was used as primary method of analysis.
Time Frame: At Weeks 56, 76, 100 and 148
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | DTG + RPV
Number analyzed (Participants) | 257
Score on a scale
  Total score, Week 56 | 0.0 [-37 to 26]
  Total score, Week 76 | 1.0 [-35 to 26]
  Total score, Week 100 | 0.0 [-27 to 26]
  Total score, Week 148 | 1.0 [-38 to 26]
  lifestyle/ease Sub-score, Week 56 | 0.0 [-21 to 12]
  lifestyle/ease Sub-score, Week 76 | 0.0 [-21 to 12]
  lifestyle/ease Sub-score, Week 100 | 0.0 [-18 to 12]
  lifestyle/ease Sub-score, Week 148 | 0.0 [-18 to 12]
  General Satisfaction/CS, Week 56 | 0.0 [-16 to 14]
  General Satisfaction/CS, Week 76 | 0.0 [-15 to 14]
  General Satisfaction/CS, Week 100 | 0.0 [-15 to 14]
  General Satisfaction/CS, Week 148 | 0.0 [-26 to 14]

42. Secondary Outcome: Change From LS Baseline Treatment Satisfaction Using the HIV TSQ at Weeks 56, 76, 100 and 148-CAR Group Through Late Switch Phase
Description: The HIV TSQ is a 10-item self-reported scale that measures overall satisfaction with treatment and by specific domains e.g., convenience, flexibility. Each item is scored 0 (very dissatisfied, inconvenient) to 6 (very satisfied, convenient). The items are summed up to produce a treatment satisfaction total score (0 to 60) and 2 subscale scores: general satisfaction/clinical and lifestyle/ease subscales (0 to 30). Higher scores indicated greater treatment satisfaction as compared to the past few weeks. The HIV TSQ was administered as a paper questionnaire. Change from LS Baseline is calculated as the value at specified time point minus LS Baseline value. Total score, lifestyle/ease score and General satisfaction/CS have been summarized. LOCF was used as primary method of analysis.
Time Frame: At Weeks 56, 76, 100 and 148
Population: LS ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 239
Score on a scale
  Total score, Week 56: number analyzed (Participants) | 235
  Total score, Week 56 | 0.0 [-17 to 52]
  Total score, Week 76 | 0.0 [-26 to 52]
  Total score, Week 100 | 0.0 [-17 to 51]
  Total score, Week 148 | 0.0 [-17 to 51]
  lifestyle/ease Sub-score, Week 56: number analyzed (Participants) | 235
  lifestyle/ease Sub-score, Week 56 | 0.0 [-10 to 22]
  lifestyle/ease Sub-score, Week 76 | 0.0 [-12 to 22]
  lifestyle/ease Sub-score, Week 100 | 0.0 [-9 to 22]
  lifestyle/ease Sub-score, Week 148 | 0.0 [-10 to 22]
  General Satisfaction/CS, Week 56: number analyzed (Participants) | 235
  General Satisfaction/CS, Week 56 | 0.0 [-12 to 30]
  General Satisfaction/CS, Week 76 | 0.0 [-15 to 30]
  General Satisfaction/CS, Week 100 | 0.0 [-9 to 29]
  General Satisfaction/CS, Week 148 | 0.0 [-9 to 29]

43. Other Pre Specified Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Weeks 100 and 148 Using the Snapshot Algorithm-DTG+RPV Group Through Early and Late Switch Phase
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Percentage of participants with plasma HIV 1 RNA < 50 c/mL using the FDA snapshot algorithm was assessed. Virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment within the window of the visit of interest.
Time Frame: Weeks 100 and 148
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 261
Percentage of participants
  Week 100 | 89
  Week 148 | 84

44. Other Pre Specified Outcome: Change From Baseline in CD4+ Lymphocyte Count at Weeks 100 and 148-DTG+RPV Group Through Early and Late Switch Phase
Description: Blood samples were collected for CD4+ cell count assessment by flow cytometry. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Weeks 100 and 148
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | DTG + RPV
Number analyzed (Participants) | 261
Cells/mm^3
  Week 100: number analyzed (Participants) | 235
  Week 100 | 55.9 (202.56)
  Week 148: number analyzed (Participants) | 221
  Week 148 | 51.5 (205.98)

45. Other Pre Specified Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Weeks 100 and 148 Using the Snapshot Algorithm-CAR Group Through Late Switch Phase
Description: as for outcome 43
Time Frame: Weeks 100 and 148
Population: LS ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 239
Percentage of participants
  Week 100 | 97
  Week 148 | 93

46. Other Pre Specified Outcome: Change From LS Baseline in CD4+ Lymphocyte Count at Weeks 100 and 148-CAR Group Through Late Switch Phase
Description: Blood samples were collected for CD4+ cell count assessment by flow cytometry. Change from LS Baseline was calculated as value at indicated time point minus LS Baseline value.
Time Frame: LS Baseline (Week 48), Weeks 100 and 148
Population: LS ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 239
Cells/mm^3
  Week 100: number analyzed (Participants) | 231
  Week 100 | 20.9 (173.39)
  Week 148: number analyzed (Participants) | 225
  Week 148 | 6.5 (167.44)

47. Secondary Outcome: Number of Participants With Observed Genotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class-DTG+RPV Group Through Continuation Phase
Description: For all participants who met virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were analyzed in an attempt to obtain genotype data on as many samples as possible. Samples for drug resistance testing (genotypic) were collected at Day 1. Number of participants with genotypic resistance to DTG or RPV for those meeting virologic withdrawal criteria in subgroups, stratified based on baseline third agent treatment class (NNRTI) were summarized.
Time Frame: Up to Week 410
Population: The analysis was performed on the CVW Resistance population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 2
Participants
  NNRTI, INI, DTG, Susceptible | 2
  NNRTI, INI, DTG, Potential low-level resistance | 0
  NNRTI, INI, DTG, Low-level resistance | 0
  NNRTI, INI, DTG, Intermediate resistance | 0
  NNRTI, INI, DTG, High-level resistance | 0
  NNRTI, INI, EVG, Susceptible | 2
  NNRTI, INI, EVG, Potential low-level resistance | 0
  NNRTI, INI, EVG, Low-level resistance | 0
  NNRTI, INI, EVG, Intermediate resistance | 0
  NNRTI, INI, EVG, High-level resistance | 0
  NNRTI, INI, RAL, Susceptible | 2
  NNRTI, INI, RAL, Potential low-level resistance | 0
  NNRTI, INI, RAL, Low-level resistance | 0
  NNRTI, INI, RAL, Intermediate resistance | 0
  NNRTI, INI, RAL, High-level resistance | 0
  NNRTI, NNRTI, DLV, Susceptible | 2
  NNRTI, NNRTI, DLV, Potential low-level resistance | 0
  NNRTI, NNRTI, DLV, Low-level resistance | 0
  NNRTI, NNRTI, DLV, Intermediate resistance | 0
  NNRTI, NNRTI, DLV, High-level resistance | 0
  NNRTI, NNRTI, EFV, Susceptible | 0
  NNRTI, NNRTI, EFV, Potential low-level resistance | 0
  NNRTI, NNRTI, EFV, Low-level resistance | 1
  NNRTI, NNRTI, EFV, Intermediate resistance | 0
  NNRTI, NNRTI, EFV, High-level resistance | 1
  NNRTI, NNRTI, ETR, Susceptible | 0
  NNRTI, NNRTI, ETR, Potential low-level resistance | 0
  NNRTI, NNRTI, ETR, Low-level resistance | 1
  NNRTI, NNRTI, ETR, Intermediate resistance | 0
  NNRTI, NNRTI, ETR, High-level resistance | 1
  NNRTI, NNRTI, NVF, Susceptible | 0
  NNRTI, NNRTI, NVF, Potential low-level resistance | 0
  NNRTI, NNRTI, NVF, Low-level resistance | 0
  NNRTI, NNRTI, NVF, Intermediate resistance | 1
  NNRTI, NNRTI, NVF, High-level resistance | 1
  NNRTI, NNRTI, RPV, Susceptible | 0
  NNRTI, NNRTI, RPV, Potential low-level resistance | 0
  NNRTI, NNRTI, RPV, Low-level resistance | 0
  NNRTI, NNRTI, RPV, Intermediate resistance | 1
  NNRTI, NNRTI, RPV, High-level resistance | 1
  NNRTI, NRTI, 3TC, Susceptible | 0
  NNRTI, NRTI, 3TC, Potential low-level resistance | 0
  NNRTI, NRTI, 3TC, Low-level resistance | 0
  NNRTI, NRTI, 3TC, Intermediate resistance | 0
  NNRTI, NRTI, 3TC, High-level resistance | 0
  NNRTI, NRTI, ABC, Susceptible | 2
  NNRTI, NRTI, ABC, Potential low-level resistance | 0
  NNRTI, NRTI, ABC, Low-level resistance | 0
  NNRTI, NRTI, ABC, Intermediate resistance | 0
  NNRTI, NRTI, ABC, High-level resistance | 0
  NNRTI, NRTI, FTC, Susceptible | 2
  NNRTI, NRTI, FTC, Potential low-level resistance | 0
  NNRTI, NRTI, FTC, Low-level resistance | 0
  NNRTI, NRTI, FTC, Intermediate resistance | 0
  NNRTI, NRTI, FTC, High-level resistance | 0
  NNRTI, NRTI, TDF, Susceptible | 2
  NNRTI, NRTI, TDF, Potential low-level resistance | 0
  NNRTI, NRTI, TDF, Low-level resistance | 0
  NNRTI, NRTI, TDF, Intermediate resistance | 0
  NNRTI, NRTI, TDF, High-level resistance | 0
  NNRTI, NRTI, ZDF, Susceptible | 2
  NNRTI, NRTI, ZDF, Potential low-level resistance | 0
  NNRTI, NRTI, ZDF, Low-level resistance | 0
  NNRTI, NRTI, ZDF, Intermediate resistance | 0
  NNRTI, NRTI, ZDF, High-level resistance | 0
  NNRTI, NRTI, d4T, Susceptible | 2
  NNRTI, NRTI, d4T, Potential low-level resistance | 0
  NNRTI, NRTI, d4T, Low-level resistance | 0
  NNRTI, NRTI, d4T, Intermediate resistance | 0
  NNRTI, NRTI, d4T, High-level resistance | 0
  NNRTI, PI, ATV/r, Susceptible | 2
  NNRTI, PI, ATV/r, Potential low-level resistance | 0
  NNRTI, PI, ATV/r, Low-level resistance | 0
  NNRTI, PI, ATV/r, Intermediate resistance | 0
  NNRTI, PI, ATV/r, High-level resistance | 0
  NNRTI, PI, DRV/r, Susceptible | 2
  NNRTI, PI, DRV/r, Potential low-level resistance | 0
  NNRTI, PI, DRV/r, Low-level resistance | 0
  NNRTI, PI, DRV/r, Intermediate resistance | 0
  NNRTI, PI, DRV/r, High-level resistance | 0
  NNRTI, PI, FPV/r, Susceptible | 2
  NNRTI, PI, FPV/r, Potential low-level resistance | 0
  NNRTI, PI, FPV/r, Low-level resistance | 0
  NNRTI, PI, FPV/r, Intermediate resistance | 0
  NNRTI, PI, FPV/r, High-level resistance | 0
  NNRTI, PI, IDV/r, Susceptible | 2
  NNRTI, PI, IDV/r, Potential low-level resistance | 0
  NNRTI, PI, IDV/r, Low-level resistance | 0
  NNRTI, PI, IDV/r, Intermediate resistance | 0
  NNRTI, PI, IDV/r, High-level resistance | 0
  NNRTI, PI, LPV/r, Susceptible | 2
  NNRTI, PI, LPV/r, Potential low-level resistance | 0
  NNRTI, PI, LPV/r, Low-level resistance | 0
  NNRTI, PI, LPV/r, Intermediate resistance | 0
  NNRTI, PI, LPV/r, High-level resistance | 0
  NNRTI, PI, NFV, Susceptible | 2
  NNRTI, PI, NFV, Potential low-level resistance | 0
  NNRTI, PI, NFV, Low-level resistance | 0
  NNRTI, PI, NFV, Intermediate resistance | 0
  NNRTI, PI, NFV, High-level resistance | 0
  NNRTI, PI, RTV, Susceptible | 2
  NNRTI, PI, RTV, Potential low-level resistance | 0
  NNRTI, PI, RTV, Low-level resistance | 0
  NNRTI, PI, RTV, Intermediate resistance | 0
  NNRTI, PI, RTV, High-level resistance | 0
  NNRTI, PI, SQV/r, Susceptible | 2
  NNRTI, PI, SQV/r, Potential low-level resistance | 0
  NNRTI, PI, SQV/r, Low-level resistance | 0
  NNRTI, PI, SQV/r, Intermediate resistance | 0
  NNRTI, PI, SQV/r, High-level resistance | 0
  NNRTI, PI, TPV/r, Susceptible | 2
  NNRTI, PI, TPV/r, Potential low-level resistance | 0
  NNRTI, PI, TPV/r, Low-level resistance | 0
  NNRTI, PI, TPV/r, Intermediate resistance | 0
  NNRTI, PI, TPV/r, High-level resistance | 0

48. Secondary Outcome: Number of Participants With Observed Phenotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class-DTG+RPV Group Through Continuation Phase
Description: For all participants who met virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were analyzed in an attempt to obtain phenotype data on as many samples as possible. Samples for drug resistance testing (phenotypic) were collected at Day 1. Number of participants with phenotypic resistance to DTG or RPV for those meeting virologic withdrawal criteria in subgroups, stratified based on baseline third agent treatment class (NNRTI) were summarized.
Time Frame: Up to Week 410
Population: The analysis was performed on the CVW Resistance population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 2
Participants
  NNRTI, INI, DTG, Resistant: number analyzed (Participants) | 1
  NNRTI, INI, DTG, Resistant | 0
  NNRTI, INI, DTG, Partially Sensitive: number analyzed (Participants) | 1
  NNRTI, INI, DTG, Partially Sensitive | 0
  NNRTI, INI, DTG, Sensitive: number analyzed (Participants) | 1
  NNRTI, INI, DTG, Sensitive | 1
  NNRTI, INI, EVG, Resistant: number analyzed (Participants) | 1
  NNRTI, INI, EVG, Resistant | 0
  NNRTI, INI, EVG, Partially Sensitive: number analyzed (Participants) | 1
  NNRTI, INI, EVG, Partially Sensitive | 0
  NNRTI, INI, EVG, Sensitive: number analyzed (Participants) | 1
  NNRTI, INI, EVG, Sensitive | 1
  NNRTI, INI, RAL, Resistant: number analyzed (Participants) | 1
  NNRTI, INI, RAL, Resistant | 1
  NNRTI, INI, RAL, Partially Sensitive: number analyzed (Participants) | 1
  NNRTI, INI, RAL, Partially Sensitive | 0
  NNRTI, INI, RAL, Sensitive: number analyzed (Participants) | 1
  NNRTI, INI, RAL, Sensitive | 0
  NNRTI, NNRTI, DLV, Resistant | 1
  NNRTI, NNRTI, DLV, Partially Sensitive | 0
  NNRTI, NNRTI, DLV, Sensitive | 1
  NNRTI, NNRTI, EFV, Resistant | 1
  NNRTI, NNRTI, EFV, Partially Sensitive | 0
  NNRTI, NNRTI, EFV, Sensitive | 1
  NNRTI, NNRTI, ETR, Resistant | 1
  NNRTI, NNRTI, ETR, Partially Sensitive | 0
  NNRTI, NNRTI, ETR, Sensitive | 1
  NNRTI, NNRTI, NVP, Resistant: number analyzed (Participants) | 1
  NNRTI, NNRTI, NVP, Resistant | 0
  NNRTI, NNRTI, NVP, Partially Sensitive | 0
  NNRTI, NNRTI, NVP, Sensitive | 1
  NNRTI, NNRTI, RPV, Resistant | 1
  NNRTI, NNRTI, RPV, Partially Sensitive | 0
  NNRTI, NNRTI, RPV, Sensitive | 1
  NNRTI, NRTI, 3TC, Reistant | 0
  NNRTI, NRTI, 3TC, Partially Sensitive | 0
  NNRTI, NRTI, 3TC, Sensitive | 2
  NNRTI, NRTI, ABC, Resistant | 0
  NNRTI, NRTI, ABC, Partially Sensitive | 0
  NNRTI, NRTI, ABC, Sensitive | 2
  NNRTI, NRTI, FTC, Resistant | 0
  NNRTI, NRTI, FTC, Partially Sensitive | 0
  NNRTI, NRTI, FTC, Sensitive | 2
  NNRTI, NRTI, TDF, Resistant | 0
  NNRTI, NRTI, TDF, Partially Sensitive | 0
  NNRTI, NRTI, TDF, Sensitive | 2
  NNRTI, NRTI, ZDF, Resistant | 0
  NNRTI, NRTI, ZDF, Partially Sensitive | 0
  NNRTI, NRTI, ZDF, Sensitive | 2
  NNRTI, NRTI, d4T, Resistant | 0
  NNRTI, NRTI, d4T, Partially Sensitive | 0
  NNRTI, NRTI, d4T, Sensitive | 2
  NNRTI, NRTI, ddI, Resistant | 0
  NNRTI, NRTI, ddI, Partially Sensitive | 0
  NNRTI, NRTI, ddI, Sensitive | 2
  NNRTI, PI, ATV/r, Resistant | 0
  NNRTI, PI, ATV/r, Partially Sensitive | 0
  NNRTI, PI, ATV/r, Sensitive | 2
  NNRTI, PI, DRV/r, Resistant | 0
  NNRTI, PI, DRV/r, Partially Sensitive | 0
  NNRTI, PI, DRV/r, Sensitive | 2
  NNRTI, PI, FPV/r, Resistant | 0
  NNRTI, PI, FPV/r, Partially Sensitive | 0
  NNRTI, PI, FPV/r, Sensitive | 2
  NNRTI, PI, IDV/r, Resistant | 0
  NNRTI, PI, IDV/r, Partially Sensitive | 0
  NNRTI, PI, IDV/r, Sensitive | 2
  NNRTI, PI, LPV/r, yResistant | 0
  NNRTI, PI, LPV/r, Partially Sensitive | 0
  NNRTI, PI, LPV/r, Sensitive | 2
  NNRTI, PI, NFV, Resistant | 0
  NNRTI, PI, NFV, Partially Sensitive | 0
  NNRTI, PI, NFV, Sensitive | 2
  NNRTI, PI, RTV, Resistant | 0
  NNRTI, PI, RTV, Partially Sensitive | 0
  NNRTI, PI, RTV, Sensitive | 2
  NNRTI, PI, SQV/r, Resistant | 0
  NNRTI, PI, SQV/r, Partiallly Sensitive | 0
  NNRTI, PI, SQV/r, Sensitive | 2
  NNRTI, PI, TPV/r, Resistant | 0
  NNRTI, PI, TPV/r, Partially Sensitive | 0
  NNRTI, PI, TPV/r, Sensitive | 2

49. Secondary Outcome: Number of Participants With Observed Genotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class CAR Group Through Continuation Phase
Description: For all participants who meet virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were analyzed in an attempt to obtain genotype data on as many samples as possible. Number of participants with genotypic resistance to CAR for those meeting virologic withdrawal criteria in subgroups, stratified based on baseline third agent treatment class (NNRTI) were summarized.
Time Frame: Week 52 to Week 410
Population: The analysis was performed on the Late Switch CVW Resistance population.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1
Participants
  NNRTI, INI, DTG, Susceptible | 1
  NNRTI, INI, DTG, Potential low-level resistance | 0
  NNRTI, INI, DTG, Low-level resistance | 0
  NNRTI, INI, DTG, Intermediate resistance | 0
  NNRTI, INI, DTG, High-level resistance | 0
  NNRTI, INI, EVG, Susceptible | 1
  NNRTI, INI, EVG, Potential low-level resistance | 0
  NNRTI, INI, EVG, Low-level resistance | 0
  NNRTI, INI, EVG, Intermediate resistance | 0
  NNRTI, INI, EVG, High-level resistance | 0
  NNRTI, INI, RAL, Susceptible | 1
  NNRTI, INI, RAL, Potential low-level resistance | 0
  NNRTI, INI, RAL, Low-level resistance | 0
  NNRTI, INI, RAL, Intermediate resistance | 0
  NNRTI, INI, RAL, High-level resistance | 0
  NNRTI, NNRTI, DLV, Susceptible | 1
  NNRTI, NNRTI, DLV, Potential low-level resistance | 0
  NNRTI, NNRTI, DLV, Low-level resistance | 0
  NNRTI, NNRTI, DLV, Intermediate resistance | 0
  NNRTI, NNRTI, DLV, High-level resistance | 0
  NNRTI, NNRTI, EFV, Susceptible | 0
  NNRTI, NNRTI, EFV, Potential low-level resistance | 0
  NNRTI, NNRTI, EFV, Low-level resistance | 0
  NNRTI, NNRTI, EFV, Intermediate resistance | 0
  NNRTI, NNRTI, EFV, High-level resistance | 1
  NNRTI, NNRTI, ETR, Susceptible | 0
  NNRTI, NNRTI, ETR, Potential low-level resistance | 0
  NNRTI, NNRTI, ETR, Low-level resistance | 0
  NNRTI, NNRTI, ETR, Intermediate resistance | 1
  NNRTI, NNRTI, ETR, High-level resistance | 0
  NNRTI, NNRTI, RPV, Susceptible | 0
  NNRTI, NNRTI, RPV, Potential low-level resistance | 0
  NNRTI, NNRTI, RPV, Low-level resistance | 0
  NNRTI, NNRTI, RPV, Intermediate resistance | 0
  NNRTI, NNRTI, RPV, High-level resistance | 1
  NNRTI, NRTI, 3TC, Susceptible | 0
  NNRTI, NRTI, 3TC, Potential low-level resistance | 0
  NNRTI, NRTI, 3TC, Low-level resistance | 0
  NNRTI, NRTI, 3TC, Intermediate resistance | 0
  NNRTI, NRTI, 3TC, High-level resistance | 0
  NNRTI, NRTI, ABC, Susceptible | 1
  NNRTI, NRTI, ABC, Potential low-level resistance | 0
  NNRTI, NRTI, ABC, Low-level resistance | 0
  NNRTI, NRTI, ABC, Intermediate resistance | 0
  NNRTI, NRTI, ABC, High-level resistance | 0
  NNRTI, NRTI, FTC, Susceptible | 1
  NNRTI, NRTI, FTC, Potential low-level resistance | 0
  NNRTI, NRTI, FTC, Low-level resistance | 0
  NNRTI, NRTI, FTC, Intermediate resistance | 0
  NNRTI, NRTI, FTC, High-level resistance | 0
  NNRTI, NRTI, TDF, Susceptible | 1
  NNRTI, NRTI, TDF, Potential low-level resistance | 0
  NNRTI, NRTI, TDF, Low-level resistance | 0
  NNRTI, NRTI, TDF, Intermediate resistance | 0
  NNRTI, NRTI, TDF, High-level resistance | 0
  NNRTI, NRTI, ZDF, Susceptible | 1
  NNRTI, NRTI, ZDF, Potential low-level resistance | 0
  NNRTI, NRTI, ZDF, Low-level resistance | 0
  NNRTI, NRTI, ZDF, Intermediate resistance | 0
  NNRTI, NRTI, ZDF, High-level resistance | 0
  NNRTI, NRTI, d4T, Susceptible | 1
  NNRTI, NRTI, d4T, Potential low-level resistance | 0
  NNRTI, NRTI, d4T, Low-level resistance | 0
  NNRTI, NRTI, d4T, Intermediate resistance | 0
  NNRTI, NRTI, d4T, High-level resistance | 0
  NNRTI, PI, ATV/r, Susceptible | 1
  NNRTI, PI, ATV/r, Potential low-level resistance | 0
  NNRTI, PI, ATV/r, Low-level resistance | 0
  NNRTI, PI, ATV/r, Intermediate resistance | 0
  NNRTI, PI, ATV/r, High-level resistance | 0
  NNRTI, PI, DRV/r, Susceptible | 1
  NNRTI, PI, DRV/r, Potential low-level resistance | 0
  NNRTI, PI, DRV/r, Low-level resistance | 0
  NNRTI, PI, DRV/r, Intermediate resistance | 0
  NNRTI, PI, DRV/r, High-level resistance | 0
  NNRTI, PI, FPV/r, Susceptible | 1
  NNRTI, PI, FPV/r, Potential low-level resistance | 0
  NNRTI, PI, FPV/r, Low-level resistance | 0
  NNRTI, PI, FPV/r, Intermediate resistance | 0
  NNRTI, PI, FPV/r, High-level resistance | 0
  NNRTI, PI, IDV/r, Susceptible | 1
  NNRTI, PI, IDV/r, Potential low-level resistance | 0
  NNRTI, PI, IDV/r, Low-level resistance | 0
  NNRTI, PI, IDV/r, Intermediate resistance | 0
  NNRTI, PI, IDV/r, High-level resistance | 0
  NNRTI, PI, LPV/r, Susceptible | 1
  NNRTI, PI, LPV/r, Potential low-level resistance | 0
  NNRTI, PI, LPV/r, Low-level resistance | 0
  NNRTI, PI, LPV/r, Intermediate resistance | 0
  NNRTI, PI, LPV/r, High-level resistance | 0
  NNRTI, PI, NFV, Susceptible | 1
  NNRTI, PI, NFV, Potential low-level resistance | 0
  NNRTI, PI, NFV, Low-level resistance | 0
  NNRTI, PI, NFV, Intermediate resistance | 0
  NNRTI, PI, NFV, High-level resistance | 0
  NNRTI, PI, RTV, Susceptible | 1
  NNRTI, PI, RTV, Potential low-level resistance | 0
  NNRTI, PI, RTV, Low-level resistance | 0
  NNRTI, PI, RTV, Intermediate resistance | 0
  NNRTI, PI, RTV, High-level resistance | 0
  NNRTI, PI, SQV/r, Susceptible | 1
  NNRTI, PI, SQV/r, Potential low-level resistance | 0
  NNRTI, PI, SQV/r, Low-level resistance | 0
  NNRTI, PI, SQV/r, Intermediate resistance | 0
  NNRTI, PI, SQV/r, High-level resistance | 0
  NNRTI, PI, TPV/r, Susceptible | 1
  NNRTI, PI, TPV/r, Potential low-level resistance | 0
  NNRTI, PI, TPV/r, Low-level resistance | 0
  NNRTI, PI, TPV/r, Intermediate resistance | 0
  NNRTI, PI, TPV/r, High-level resistance | 0
  NNRTI, NNRTI, NVP, Susceptible | 0
  NNRTI, NNRTI, NCP, Potential low-level resistance | 0
  NNRTI, NNRTI, NVP, Low-level resistance | 0
  NNRTI, NNRTI, NVP, Intermediate resistance | 0
  NNRTI, NNRTI, NVP, High-level resistance | 1
  NNRTI, NRTI, ddI, Susceptible | 1
  NNRTI, NRTI, ddI, Potential low-level resistance | 0
  NNRTI, NRTI, ddI, Low-level resistance | 0
  NNRTI, NRTI, ddI, Intermediate resistance | 0
  NNRTI, NRTI, ddI, High-level resistance | 0

50. Secondary Outcome: Number of Participants With Observed Phenotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class- CAR Group Through Continuation Phase
Description: For all participants who meet virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were analyzed in an attempt to obtain phenotype data on as many samples as possible. Number of participants with phenotypic resistance to CAR for those meeting virologic withdrawal criteria in subgroups, stratified based on baseline third agent treatment class (NNRTI) were summarized.
Time Frame: Week 52 to Week 410
Population: The analysis was performed on the Late Switch CVW resistance population.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1
Participants
  NNRTI, NNRTI, DLV, Resistant | 1
  NNRTI, NNRTI, DLV, Partially Sensitive | 0
  NNRTI, NNRTI, DLV, Sensitive | 0
  NNRTI, NNRTI, EFV, Resistant | 1
  NNRTI, NNRTI, EFV, Partially Sensitive | 0
  NNRTI, NNRTI, EFV, Sensitive | 0
  NNRTI, NNRTI, ETR, Resistant | 0
  NNRTI, NNRTI, ETR, Partially Sensitive | 1
  NNRTI, NNRTI, ETR, Sensitive | 0
  NNRTI, NNRTI, NVP, Resistant | 1
  NNRTI, NNRTI, NVP, Partially Sensitive | 0
  NNRTI, NNRTI, NVP, Sensitive | 0
  NNRTI, NNRTI, RPV, Resistant | 1
  NNRTI, NNRTI, RPV, Partially Sensitive | 0
  NNRTI, NNRTI, RPV, Sensitive | 0
  NNRTI, NRTI, 3TC, Reistant | 0
  NNRTI, NRTI, 3TC, Partially Sensitive | 0
  NNRTI, NRTI, 3TC, Sensitive | 1
  NNRTI, NRTI, ABC, Resistant | 0
  NNRTI, NRTI, ABC, Partially Sensitive | 0
  NNRTI, NRTI, ABC, Sensitive | 1
  NNRTI, NRTI, FTC, Resistant | 0
  NNRTI, NRTI, FTC, Partially Sensitive | 0
  NNRTI, NRTI, FTC, Sensitive | 1
  NNRTI, NRTI, TDF, Resistant | 0
  NNRTI, NRTI, TDF, Partially Sensitive | 0
  NNRTI, NRTI, TDF, Sensitive | 1
  NNRTI, NRTI, ZDF, Resistant | 0
  NNRTI, NRTI, ZDF, Partially Sensitive | 0
  NNRTI, NRTI, ZDF, Sensitive | 1
  NNRTI, NRTI, d4T, Resistant | 0
  NNRTI, NRTI, d4T, Partially Sensitive | 0
  NNRTI, NRTI, d4T, Sensitive | 1
  NNRTI, NRTI, ddI, Resistant | 0
  NNRTI, NRTI, ddI, Partially Sensitive | 0
  NNRTI, NRTI, ddI, Sensitive | 1
  NNRTI, PI, ATV/r, Resistant | 0
  NNRTI, PI, ATV/r, Partially Sensitive | 0
  NNRTI, PI, ATV/r, Sensitive | 1
  NNRTI, PI, DRV/r, Resistant | 0
  NNRTI, PI, DRV/r, Partially Sensitive | 0
  NNRTI, PI, DRV/r, Sensitive | 1
  NNRTI, PI, FPV/r, Resistant | 0
  NNRTI, PI, FPV/r, Partially Sensitive | 0
  NNRTI, PI, FPV/r, Sensitive | 1
  NNRTI, PI, IDV/r, Resistant | 0
  NNRTI, PI, IDV/r, Partially Sensitive | 0
  NNRTI, PI, IDV/r, Sensitive | 1
  NNRTI, PI, LPV/r, Resistant | 0
  NNRTI, PI, LPV/r, Partially Sensitive | 0
  NNRTI, PI, LPV/r, Sensitive | 1
  NNRTI, PI, NFV, Resistant | 0
  NNRTI, PI, NFV, Partially Sensitive | 0
  NNRTI, PI, NFV, Sensitive | 1
  NNRTI, PI, RTV, Resistant | 0
  NNRTI, PI, RTV, Partially Sensitive | 0
  NNRTI, PI, RTV, Sensitive | 1
  NNRTI, PI, SQV/r, Resistant | 0
  NNRTI, PI, SQV/r, Partiallly Sensitive | 0
  NNRTI, PI, SQV/r, Sensitive | 1
  NNRTI, PI, TPV/r, Resistant | 0
  NNRTI, PI, TPV/r, Partially Sensitive | 0
  NNRTI, PI, TPV/r, Sensitive | 1

51. Secondary Outcome: Number of Participants With Genotypic Resistance-DTG+RPV Group Through Continuation Phase
Description: Plasma samples were collected for participants meeting the CVW criteria (previous plasma HIV-1 RNA >=50 c/mL and current plasma HIV-1 RNA >= 200 c/mL) to evaluate any potential genotypic evolution of resistance. Genotypic Resistance data for the following drugs was presented: DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r, TPV/r.
Time Frame: Up to Week 410
Population: The analysis was performed on the CVW Resistance population which included all participants from the Intent-to-Treat Exposed (ITT-E) population who met CVW through the end of the visit window and had available on-treatment genotypic resistance data at the time the CVW criterion was met.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 2
Participants
  INI, DTG, Susceptible | 2
  INI, DTG, Potential low-level resistance | 0
  INI, DTG, Low-level resistance | 0
  INI, DTG, Intermediate resistance | 0
  INI, DTG, High-level resistance | 0
  INI, EVG, Susceptible | 2
  INI, EVG, Potential low-level resistance | 0
  INI, EVG, Low-level resistance | 0
  INI, EVG, Intermediate resistance | 0
  INI, EVG, High-level resistance | 0
  INI, RAL, Susceptible | 2
  INI, RAL, Potential low-level resistance | 0
  INI, RAL, Low-level resistance | 0
  INI, RAL, Intermediate resistance | 0
  INI, RAL, High-level resistance | 0
  NNRTI, DLV, Susceptible | 2
  NNRTI, DLV, Potential low-level resistance | 0
  NNRTI, DLV, Low-level resistance | 0
  NNRTI, DLV, Intermediate resistance | 0
  NNRTI, DLV, High-level resistance | 0
  NNRTI, EFV, Susceptible | 0
  NNRTI, EFV, Potential low-level resistance | 0
  NNRTI, EFV, Low-level resistance | 1
  NNRTI, EFV, Intermediate resistance | 0
  NNRTI, EFV, High-level resistance | 1
  NNRTI, ETR, Susceptible | 0
  NNRTI, ETR, Potential low-level resistance | 0
  NNRTI, ETR, Low-level resistance | 1
  NNRTI, ETR, Intermediate resistance | 0
  NNRTI, ETR, High-level resistance | 1
  NNRTI, NVP, Susceptible | 0
  NNRTI, NVP, Potential low-level resistance | 0
  NNRTI, NVP, Low-level resistance | 0
  NNRTI, NVP, Intermediate resistance | 1
  NNRTI, NVP, High-level resistance | 1
  NNRTI, RPV, Susceptible | 0
  NNRTI, RPV, Potential low-level resistance | 0
  NNRTI, RPV, Low-level resistance | 0
  NNRTI, RPV, Intermediate resistance | 1
  NNRTI, RPV, High-level resistance | 1
  NRTI, 3TC, Susceptible | 2
  NRTI, 3TC, Potential low-level resistance | 0
  NRTI, 3TC, Low-level resistance | 0
  NRTI, 3TC, Intermediate resistance | 0
  NRTI, 3TC, High-level resistance | 0
  NRTI, ABC, Susceptible | 2
  NRTI, ABC, Potential low-level resistance | 0
  NRTI, ABC, Low-level resistance | 0
  NRTI, ABC, Intermediate resistance | 0
  NRTI, ABC, High-level resistance | 0
  NRTI, FTC, Susceptible | 2
  NRTI, FTC, Potential low-level resistance | 0
  NRTI, FTC, Low-level resistance | 0
  NRTI, FTC, Intermediate resistance | 0
  NRTI, FTC, High-level resistance | 0
  NRTI, TDF, Susceptible | 2
  NRTI, TDF, Potential low-level resistance | 0
  NRTI, TDF, Low-level resistance | 0
  NRTI, TDF, Intermediate resistance | 0
  NRTI, TDF, High-level resistance | 0
  NRTI, ZDV, Susceptible | 2
  NRTI, ZDV, Potential low-level resistance | 0
  NRTI, ZDV, Low-level resistance | 0
  NRTI, ZDV, Intermediate resistance | 0
  NRTI, ZDV, High-level resistance | 0
  NRTI, d4T, Susceptible | 2
  NRTI, d4T, Potential low-level resistance | 0
  NRTI, d4T, Low-level resistance | 0
  NRTI, d4T, Intermediate resistance | 0
  NRTI, d4T, High-level resistance | 0
  NRTI, ddI, Susceptible | 2
  NRTI, ddI, Potential low-level resistance | 0
  NRTI, ddI, Low-level resistance | 0
  NRTI, ddI, Intermediate resistance | 0
  NRTI, ddI, High-level resistance | 0
  PI, ATV/r, Susceptible | 2
  PI, ATV/r, Potential low-level resistance | 0
  PI, ATV/r, Low-level resistance | 0
  PI, ATV/r, Intermediate resistance | 0
  PI, ATV/r, High-level resistance | 0
  PI, DRV/r, Susceptible | 2
  PI, DRV/r, Potential low-level resistance | 0
  PI, DRV/r, Low-level resistance | 0
  PI, DRV/r, Intermediate resistance | 0
  PI, DRV/r, High-level resistance | 0
  PI, FPV/r, Susceptible | 2
  PI, FPV/r, Potential low-level resistance | 0
  PI, FPV/r, Low-level resistance | 0
  PI, FPV/r, Intermediate resistance | 0
  PI, FPV/r, High-level resistance | 0
  PI, IDV/r, Susceptible | 2
  PI, IDV/r, Potential low-level resistance | 0
  PI, IDV/r, Low-level resistance | 0
  PI, IDV/r, Intermediate resistance | 0
  PI, IDV/r, High-level resistance | 0
  PI, LPV/r, Susceptible | 2
  PI, LPV/r, Potential low-level resistance | 0
  PI, LPV/r, Low-level resistance | 0
  PI, LPV/r, Intermediate resistance | 0
  PI, LPV/r, High-level resistance | 0
  PI, NFV, Susceptible | 2
  PI, NFV, Potential low-level resistance | 0
  PI, NFV, Low-level resistance | 0
  PI, NFV, Intermediate resistance | 0
  PI, NFV, High-level resistance | 0
  PI, RTV, Susceptible | 2
  PI, RTV, Potential low-level resistance | 0
  PI, RTV, Low-level resistance | 0
  PI, RTV, Intermediate resistance | 0
  PI, RTV, High-level resistance | 0
  PI, SQV/r, Susceptible | 2
  PI, SQV/r, Potential low-level resistance | 0
  PI, SQV/r, Low-level resistance | 0
  PI, SQV/r, Intermediate resistance | 0
  PI, SQV/r, High-level resistance | 0
  PI, TPV/r, Susceptible | 2
  PI, TPV/r, Potential low-level resistance | 0
  PI, TPV/r, Low-level resistance | 0
  PI, TPV/r, Intermediate resistance | 0
  PI, TPV/r, High-level resistance | 0

52. Secondary Outcome: Number of Participants With Phenotypic Resistance-DTG+RPV Group Through Continuation Phase
Description: Plasma samples were collected for participants meeting the CVW criteria (previous plasma HIV-1 RNA >=50 c/mL and current plasma HIV-1 RNA >= 200 c/mL) to evaluate any potential phenotypic evolution of resistance. Phenotypic Resistance data for the following drugs was presented: DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r, TPV/r.
Time Frame: Up to Week 410
Population: The analysis was performed on the CVW Resistance population which included all participants from the ITT-E population who met CVW through the end of the visit window and had available on-treatment phenotypic resistance data at the time the CVW criterion was met.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 2
Participants
  INI, DTG, Resistant | 0
  INI, DTG, Partially Sensitive | 0
  INI, DTG, Sensitive | 1
  INI, EVG, Resistant | 0
  INI, EVG, Partially Sensitive | 0
  INI, EVG, Sensitive | 1
  INI, RAL, Resistant | 1
  INI, RAL, Partially Sensitive | 0
  INI, RAL, Sensitive | 0
  NNRTI, DLV, Resistant | 1
  NNRTI, DLV, Partially Sensitive | 0
  NNRTI, DLV, Sensitive | 1
  NNRTI, EFV, Resistant | 1
  NNRTI, EFV, Partially Sensitive | 0
  NNRTI, EFV, Sensitive | 1
  NNRTI, ETR, Resistant | 1
  NNRTI, ETR, Partially Sensitive | 0
  NNRTI, ETR, Sensitive | 1
  NNRTI, NVP, Resistant | 1
  NNRTI, NVP, Partially Sensitive | 0
  NNRTI, NVP, Sensitive | 1
  NNRTI, RPV, Resistant | 1
  NNRTI, RPV, Partially Sensitive | 0
  NNRTI, RPV, Sensitive | 1
  NRTI, 3TC, Resistant | 0
  NRTI, 3TC, Partially Sensitive | 0
  NRTI, 3TC, Sensitive | 2
  NRTI, ABC, Resistant | 0
  NRTI, ABC, Partially Sensitive | 0
  NRTI, ABC, Sensitive | 2
  NRTI, FTC, Resistant | 0
  NRTI, FTC, Partially Sensitive | 0
  NRTI, FTC, Sensitive | 2
  NRTI, TDF, Resistant | 0
  NRTI, TDF, Partially Sensitive | 0
  NRTI, TDF, Sensitive | 2
  NRTI, ZDV, Resistant | 0
  NRTI, ZDV, Partially Sensitive | 0
  NRTI, ZDV, Sensitive | 2
  NRTI, d4T, Resistant | 0
  NRTI, d4T, Partially Sensitive | 0
  NRTI, d4T, Sensitive | 2
  NRTI, ddI, Resistant | 0
  NRTI, ddI, Partially Sensitive | 0
  NRTI, ddI, Sensitive | 2
  PI, ATV/r, Resistant | 0
  PI, ATV/r, Partially Sensitive | 0
  PI, ATV/r, Sensitive | 2
  PI, DRV/r, Resistant | 0
  PI, DRV/r, Partially Sensitive | 0
  PI, DRV/r, Sensitive | 2
  PI, FPV/r, Resistant | 0
  PI, FPV/r, Partially Sensitive | 0
  PI, FPV/r, Sensitive | 2
  PI, IDV/r, Resistant | 0
  PI, IDV/r, Partially Sensitive | 0
  PI, IDV/r, Sensitive | 2
  PI, LPV/r, Resistant | 0
  PI, LPV/r, Partially Sensitive | 0
  PI, LPV/r, Sensitive | 2
  PI, NFV, Resistant | 0
  PI, NFV, Partially Sensitive | 0
  PI, NFV, Sensitive | 2
  PI, RTV, Resistant | 0
  PI, RTV, Partially Sensitive | 0
  PI, RTV, Sensitive | 2
  PI, SQV/r, Resistant | 0
  PI, SQV/r, Partially Sensitive | 0
  PI, SQV/r, Sensitive | 2
  PI, TPV/r, Resistant | 0
  PI, TPV/r, Partially Sensitive | 0
  PI, TPV/r, Sensitive | 2

53. Secondary Outcome: Number of Participants With Genotypic Resistance-CAR Group Through Continuation Phase
Description: as for outcome 52
Time Frame: Week 52 to Week 410
Population: The analysis was performed on the Late Switch CVW resistance population which included all participants from the Late Switch ITT-E population who met CVW through the end of visit window and had available on-treatment genotypic resistance data at the time the CVW criterion was met.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1
Participants
  INI, DTG, Susceptible | 1
  INI, DTG, Potential low-level resistance | 0
  INI, DTG, Low-level resistance | 0
  INI, DTG, Intermediate resistance | 0
  INI, DTG, High-level resistance | 0
  INI, EVG, Susceptible | 1
  INI, EVG, Potential low-level resistance | 0
  INI, EVG, Low-level resistance | 0
  INI, EVG, Intermediate resistance | 0
  INI, EVG, High-level resistance | 0
  INI, RAL, Susceptible | 1
  INI, RAL, Potential low-level resistance | 0
  INI, RAL, Low-level resistance | 0
  INI, RAL, Intermediate resistance | 0
  INI, RAL, High-level resistance | 0
  NNRTI, DLV, Susceptible | 1
  NNRTI, DLV, Potential low-level resistance | 0
  NNRTI, DLV, Low-level resistance | 0
  NNRTI, DLV, Intermediate resistance | 0
  NNRTI, DLV, High-level resistance | 0
  NNRTI, EFV, Susceptible | 0
  NNRTI, EFV, Potential low-level resistance | 0
  NNRTI, EFV, Low-level resistance | 0
  NNRTI, EFV, Intermediate resistance | 0
  NNRTI, EFV, High-level resistance | 1
  NNRTI, ETR, Susceptible | 0
  NNRTI, ETR, Potential low-level resistance | 0
  NNRTI, ETR, Low-level resistance | 0
  NNRTI, ETR, Intermediate resistance | 1
  NNRTI, ETR, High-level resistance | 0
  NNRTI, NVP, Susceptible | 0
  NNRTI, NVP, Potential low-level resistance | 0
  NNRTI, NVP, Low-level resistance | 0
  NNRTI, NVP, Intermediate resistance | 0
  NNRTI, NVP, High-level resistance | 1
  NNRTI, RPV, Susceptible | 0
  NNRTI, RPV, Potential low-level resistance | 0
  NNRTI, RPV, Low-level resistance | 0
  NNRTI, RPV, Intermediate resistance | 0
  NNRTI, RPV, High-level resistance | 1
  NRTI, 3TC, Susceptible | 1
  NRTI, 3TC, Potential low-level resistance | 0
  NRTI, 3TC, Low-level resistance | 0
  NRTI, 3TC, Intermediate resistance | 0
  NRTI, 3TC, High-level resistance | 0
  NRTI, ABC, Susceptible | 1
  NRTI, ABC, Potential low-level resistance | 0
  NRTI, ABC, Low-level resistance | 0
  NRTI, ABC, Intermediate resistance | 0
  NRTI, ABC, High-level resistance | 0
  NRTI, FTC, Susceptible | 1
  NRTI, FTC, Potential low-level resistance | 0
  NRTI, FTC, Low-level resistance | 0
  NRTI, FTC, Intermediate resistance | 0
  NRTI, FTC, High-level resistance | 0
  NRTI, TDF, Susceptible | 1
  NRTI, TDF, Potential low-level resistance | 0
  NRTI, TDF, Low-level resistance | 0
  NRTI, TDF, Intermediate resistance | 0
  NRTI, TDF, High-level resistance | 0
  NRTI, ZDV, Susceptible | 1
  NRTI, ZDV, Potential low-level resistance | 0
  NRTI, ZDV, Low-level resistance | 0
  NRTI, ZDV, Intermediate resistance | 0
  NRTI, ZDV, High-level resistance | 0
  NRTI, d4T, Susceptible | 1
  NRTI, d4T, Potential low-level resistance | 0
  NRTI, d4T, Low-level resistance | 0
  NRTI, d4T, Intermediate resistance | 0
  NRTI, d4T, High-level resistance | 0
  NRTI, ddI, Susceptible | 1
  NRTI, ddI, Potential low-level resistance | 0
  NRTI, ddI, Low-level resistance | 0
  NRTI, ddI, Intermediate resistance | 0
  NRTI, ddI, High-level resistance | 0
  PI, ATV/r, Susceptible | 1
  PI, ATV/r, Potential low-level resistance | 0
  PI, ATV/r, Low-level resistance | 0
  PI, ATV/r, Intermediate resistance | 0
  PI, ATV/r, High-level resistance | 0
  PI, DRV/r, Susceptible | 1
  PI, DRV/r, Potential low-level resistance | 0
  PI, DRV/r, Low-level resistance | 0
  PI, DRV/r, Intermediate resistance | 0
  PI, DRV/r, High-level resistance | 0
  PI, FPV/r, Susceptible | 1
  PI, FPV/r, Potential low-level resistance | 0
  PI, FPV/r, Low-level resistance | 0
  PI, FPV/r, Intermediate resistance | 0
  PI, FPV/r, High-level resistance | 0
  PI, IDV/r, Susceptible | 1
  PI, IDV/r, Potential low-level resistance | 0
  PI, IDV/r, Low-level resistance | 0
  PI, IDV/r, Intermediate resistance | 0
  PI, IDV/r, High-level resistance | 0
  PI, LPV/r, Susceptible | 1
  PI, LPV/r, Potential low-level resistance | 0
  PI, LPV/r, Low-level resistance | 0
  PI, LPV/r, Intermediate resistance | 0
  PI, LPV/r, High-level resistance | 0
  PI, NFV, Susceptible | 1
  PI, NFV, Potential low-level resistance | 0
  PI, NFV, Low-level resistance | 0
  PI, NFV, Intermediate resistance | 0
  PI, NFV, High-level resistance | 0
  PI, RTV, Susceptible | 1
  PI, RTV, Potential low-level resistance | 0
  PI, RTV, Low-level resistance | 0
  PI, RTV, Intermediate resistance | 0
  PI, RTV, High-level resistance | 0
  PI, SQV/r, Susceptible | 1
  PI, SQV/r, Potential low-level resistance | 0
  PI, SQV/r, Low-level resistance | 0
  PI, SQV/r, Intermediate resistance | 0
  PI, SQV/r, High-level resistance | 0
  PI, TPV/r, Susceptible | 1
  PI, TPV/r, Potential low-level resistance | 0
  PI, TPV/r, Low-level resistance | 0
  PI, TPV/r, Intermediate resistance | 0
  PI, TPV/r, High-level resistance | 0

54. Secondary Outcome: Number of Participants With Phenotypic Resistance- CAR Group Through Continuation Phase
Description: Plasma samples were collected for participants meeting the CVW criteria (previous plasma HIV-1 RNA >=50 c/mL and current plasma HIV-1 RNA >= 200 c/mL) to evaluate any potential phenotypic evolution of resistance. Phenotypic resistance data for the following drugs was presented: DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r, TPV/r.
Time Frame: Week 52 to Week 410
Population: The analysis was performed on the Late Switch CVW Resistance population which included all participants from the Late Switch ITT-E population who met CVW through the end of visit window and had available on-treatment phenotypic resistance data at the time the CVW criterion was met.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1
Participants
  NNRTI, DLV, Resistant | 1
  NNRTI, DLV, Partially Sensitive | 0
  NNRTI, DLV, Sensitive | 0
  NNRTI, EFV, Resistant | 1
  NNRTI, EFV, Partially Sensitive | 0
  NNRTI, EFV, Sensitive | 0
  NNRTI, ETR, Resistant | 0
  NNRTI, ETR, Partially Sensitive | 1
  NNRTI, ETR, Sensitive | 0
  NNRTI, NVP, Resistant | 1
  NNRTI, NVP, Partially Sensitive | 0
  NNRTI, NVP, Sensitive | 0
  NNRTI, RPV, Resistant | 1
  NNRTI, RPV, Partially Sensitive | 0
  NNRTI, RPV, Sensitive | 0
  NRTI, 3TC, Resistant | 0
  NRTI, 3TC, Partially Sensitive | 0
  NRTI, 3TC, Sensitive | 1
  NRTI, ABC, Resistant | 0
  NRTI, ABC, Partially Sensitive | 0
  NRTI, ABC, Sensitive | 1
  NRTI, FTC, Resistant | 0
  NRTI, FTC, Partially Sensitive | 0
  NRTI, FTC, Sensitive | 1
  NRTI, TDF, Resistant | 0
  NRTI, TDF, Partially Sensitive | 0
  NRTI, TDF, Sensitive | 1
  NRTI, ZDV, Resistant | 0
  NRTI, ZDV, Partially Sensitive | 0
  NRTI, ZDV, Sensitive | 1
  NRTI, d4T, Resistant | 0
  NRTI, d4T, Partially Sensitive | 0
  NRTI, d4T, Sensitive | 1
  NRTI, ddI, Resistant | 0
  NRTI, ddI, Partially Sensitive | 0
  NRTI, ddI, Sensitive | 1
  PI, ATV/r, Resistant | 0
  PI, ATV/r, Partially Sensitive | 0
  PI, ATV/r, Sensitive | 1
  PI, DRV/r, Resistant | 0
  PI, DRV/r, Partially Sensitive | 0
  PI, DRV/r, Sensitive | 1
  PI, FPV/r, Resistant | 0
  PI, FPV/r, Partially Sensitive | 0
  PI, FPV/r, Sensitive | 1
  PI, IDV/r, Resistant | 0
  PI, IDV/r, Partially Sensitive | 0
  PI, IDV/r, Sensitive | 1
  PI, LPV/r, Resistant | 0
  PI, LPV/r, Partially Sensitive | 0
  PI, LPV/r, Sensitive | 1
  PI, NFV, Resistant | 0
  PI, NFV, Partially Sensitive | 0
  PI, NFV, Sensitive | 1
  PI, RTV, Resistant | 0
  PI, RTV, Partially Sensitive | 0
  PI, RTV, Sensitive | 1
  PI, SQV/r, Resistant | 0
  PI, SQV/r, Partially Sensitive | 0
  PI, SQV/r, Sensitive | 1
  PI, TPV/r, Resistant | 0
  PI, TPV/r, Partially Sensitive | 0
  PI, TPV/r, Sensitive | 1

ADVERSE EVENTS:
Time Frame: Non-serious AEs were collected from study start until Week 148, thereafter SAEs and only AEs leading to withdrawal were collected from study start until Week 410.
Description: On treatment SAEs and non-serious AEs were reported for the Safety Population for DTG+RPV (Early Switch), CAR (Early Switch) and DTG+RPV (Early+Late Switch). LS Safety Population was used for CAR (Late Switch arm). CP Safety Population was used for DTG+RPV (Continuation Phase) and CAR (Continuation Phase).
Groups:
- DTG + RPV (Early Switch): Participants received DTG 50 mg + RPV 25 mg together once daily at approximately the same time, with a meal, in an open-label fashion up to Week 52 during early switch phase.
- CAR (Early Switch): Participants continued to receive their current antiretroviral regimen (two NRTIs + a third agent). A third agent included either an: INSTI, a NNRTI or a PI. CAR was administered according to the approved labeling in an open-label fashion up to Week 52 during early switch phase.
- DTG + RPV (Early + Late Switch): Participants received DTG 50 mg + RPV 25 mg together once daily at approximately the same time, with a meal, in an open-label fashion up to Week 52 during early switch phase. Participants continued to receive DTG 50 mg + RPV 25 mg up to Week 148 during the Late Switch Phase.
- CAR (Late Switch): Participants continued to receive their current antiretroviral regimen (two NRTIs + a third agent). A third agent included either an: INSTI, a NNRTI or a PI. CAR was administered according to the approved labeling in an open-label fashion up to Week 52 during early switch phase.
  At Week 52, participants who received CAR during the early switch phase, with HIV-1 RNA <50 c/mL, switched to DTG 50 mg + RPV 25 mg once daily and were followed until Week 148.
- DTG + RPV (Continuation Phase): Participants received DTG 50 mg + RPV 25 mg together once daily at approximately the same time, with a meal, in an open-label fashion up to Week 52 during early switch phase. Participants continued to receive DTG 50 mg + RPV 25 mg up to Week 148 during the Late Switch Phase.
  Participants who successfully completed 148 weeks of treatment were given the opportunity to continue to receive DTG + RPV once daily in the Continuation Phase (after Week 148).
- CAR (Continuation Phase): Participants continued to receive their current antiretroviral regimen (NRTIs + a third agent). A third agent included either an: INSTI, a NNRTI or a PI. CAR was administered according to the approved labeling in an open-label fashion up to Week 52 during early switch phase. At Week 52,participants with HIV-1 RNA <50 copies per milliliter (c/mL, switched to DTG 50 mg + RPV 25 mg once daily and were followed-up through the Late Switch Phase, at Week 148 and through the Continuation Phase, after Week 148.
Arm/Group | DTG + RPV (Early Switch) | CAR (Early Switch) | DTG + RPV (Early + Late Switch) | CAR (Late Switch) | DTG + RPV (Continuation Phase) | CAR (Continuation Phase)
All-Cause Mortality (participants affected / at risk) | 1/261 | 0/255 | 2/261 | 0/239 | 0/208 | 0/204
Serious Adverse Events (participants affected / at risk) | 19/261 | 9/255 | 38/261 | 22/239 | 12/208 | 12/204
Other Adverse Events (participants affected / at risk) | 121/261 | 106/255 | 170/261 | 132/239 | 0/208 | 0/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DTG + RPV (Early Switch) (N=261) | CAR (Early Switch) (N=255) | DTG + RPV (Early + Late Switch) (N=261) | CAR (Late Switch) (N=239) | DTG + RPV (Continuation Phase) (N=208) | CAR (Continuation Phase) (N=204)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic pneumonia acute (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphogranuloma venereum (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0/28 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jarisch-Herxheimer reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0/28 (0) | 0 (0)
Proctitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0/28 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Acute hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + RPV (Early Switch) (N=261) | CAR (Early Switch) (N=255) | DTG + RPV (Early + Late Switch) (N=261) | CAR (Late Switch) (N=239) | DTG + RPV (Continuation Phase) (N=208) | CAR (Continuation Phase) (N=204)
Nasopharyngitis (Infections and infestations) | 21 (26) | 23 (25) | 48 (86) | 37 (54) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 19 (21) | 27 (41) | 37 (53) | 30 (37) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 17 (20) | 11 (13) | 28 (39) | 19 (25) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (19) | 7 (7) | 25 (32) | 22 (26) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 17 (36) | 6 (6) | 27 (57) | 14 (16) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 14 (16) | 17 (23) | 22 (26) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (13) | 11 (11) | 17 (23) | 10 (12) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 6 (8) | 7 (7) | 15 (17) | 20 (24) | 0 (0) | 0 (0)
Asthenia (General disorders) | 8 (8) | 10 (11) | 14 (14) | 10 (12) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 10 (10) | 4 (5) | 19 (19) | 8 (8) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 9 (10) | 6 (6) | 16 (23) | 9 (9) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 4 (4) | 9 (9) | 13 (13) | 12 (13) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 9 (10) | 3 (4) | 18 (21) | 6 (7) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 9 (10) | 3 (3) | 15 (17) | 8 (10) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 10 (10) | 0 (0) | 14 (16) | 8 (8) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (8) | 4 (4) | 14 (17) | 7 (7) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 6 (8) | 3 (5) | 14 (16) | 4 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.